**Protocol Title:** A phase 3, open-label study to evaluate the safety of

oliceridine (TRV130) in patients with acute pain for which

parenteral opioid therapy is warranted

**Protocol Number:** CP130-3003

**Statistical Analysis Plan Version:** 1.0

**SAP Date:** 20 December 2016

**NCT:** 02656875

Client: Trevena, Inc. Version #: 1.0

Version Date: 20Dec2016

Protocol/CIP#: CP130-3003

## Protocol/CIP No. CP130-3003

A phase 3, multicenter, open-label study to evaluate the safety of oliceridine (TRV130) in patients with acute pain for which parenteral opiod therapy is warranted

## **Statistical Analysis Plan**

Prepared for:
Trevena
1018 West 8th Ave., Suite A
King of Prussia, PA 19406 USA
610-354-8840

Final Version 1.0 Date 20 December, 2016

Prepared by: Chiltern, International

## VERSION HISTORY OF IMPLEMENTED PLANS

| Version | Date | Revision Author | Comments |
|-----------|-----------|-----------------|------------------|
| Final 1.0 | 20Dec2016 | Arteid Memaj | Intitial Version |

Client: Trevena, Inc. Version #: 1.0 Version Date: 20Dec2016

Protocol/GIP#. CP130-3003

# SIGNATURE PAGE

Author:

DocuSign Envelope ID: E03C02F0-13F7-44F4-9637-A8858ECEA7AB

Arteid Memaj Biostatistician, Biometrics

200562016

Reviewed by:

Senior Wiredor, Biometrics Chiltern, International

Chiltern, International

20 Dec 2016 Date

Approved by:

-DocuSigned by: David Burt

Signer Name: David Burt Signing Reason: I approve this document Signing Time: 2016-12-21 15:24:59Z (UTC)

David Burt Director, Biostatistics Trevena, Inc.

DocuSigned by: Franck Skobieranda

Trevena, Inc.

Signer Name: Franck Skobieranda
Signing Reason: I approve this document
Signing Time: 2016-12-21 15:49:15Z (UTC)
800DD792D346408DA94BFEECB6F805C8

Vice President, Clinical Development

12/21/2016 | 10:25 EST

Date

12/21/2016 | 10:49 EST

Date


Page 2 of 30

Chiltern, International, All rights reserved. Reproduction or transmission to others apart from the parties involved with this document in any form or by any means is not permitted without the prior written consent of Chiltern, International.


Protocol/CIP#: CP130-3003

| 1. | 1 OF ABBREVIATIONS AND DEFINITIONS OF TERMS | |
|---|---|---|
| 2. | RODUCTION | 6 |
| 3. | JDY OBJECTIVES | 7 |
| 4. | UDY DESIGN | 7 |
| 4.7<br>4.7<br>4.7 | GENERAL DESIGN METHOD OF ASSIGNMENT OF PATIENTS TO CUMULATIVE DOSE GROUPS BLINDING DETERMINATION OF SAMPLE SIZE | 9<br>10 |
| 5. | ANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 10 |
| 6.<br>EVA | SELINE, SAFETY & TOLERABILITY, EFFICACY AND PHARMACOKIN | |
| 6.2<br>6.2<br>6.4 | SCHEDULE OF EVALUATIONS TIME POINT ALGORITHMS Baseline Assessments Initial Setting and Condition Category Relative Day Analysis Windows SAFETY ASSESSMENTS Extent of Exposure Adverse Events Clinical Laboratory Evaluations Vital Signs Electrocardiogram (ECG) Physical Examination Subjective Opiate Withdrawal Scale (SOWS) Oxygen Saturation Somnolence/Sedation DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETIC PARAMETERS. EFFICACY VARIABLES Numeric Pain Rating Scale (NPRS) | |
| 7. | ATISTICAL METHODS | 20 |
| 7. <sup>2</sup><br>7. <sup>2</sup><br>7. <sup>3</sup> | GENERAL METHODOLOGY ADJUSTMENTS FOR COVARIATES HANDLING OF DROPOUTS OR MISSING DATA Adverse Events Concomitant Medications Study Medication Dosing Medical History | 20<br>20<br>21 |
| | Numeric Pain Rating Scale | |


Protocol/CIP#: CP130-3003

| <i>7.3.6</i> . | Subjective Opioid Withdrawal Scale | 22 |
|----------------------|------------------------------------------------|----|
| 7.4 | INTERIM ANALYSES AND DATA MONITORING | |
| 7.5 | MULTI-CENTER STUDIES AND POOLING OF CENTERS | 22 |
| 7.6 | MULTIPLE COMPARISONS/MULTIPLICITY | 22 |
| 7.7 | EXAMINATION OF SUBGROUPS | 22 |
| 8. ST. | ATISTICAL ANALYSIS | 23 |
| 8.1 | DISPOSITION OF SUBJECTS | 23 |
| 8.2 | PROTOCOL DEVIATIONS | |
| 8.3 | ANALYSIS POPULATIONS | |
| 8.3.1. | Enrolled Analysis Set | |
| 8.3.2. | Safety Analysis Set | |
| 8.3.3. | Efficacy Analysis Set | |
| 8.4 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 8.5 | PRIOR AND CONCOMITANT MEDICATIONS | |
| 8.6 | ANALYSIS OF SAFETY | |
| 8.6.1. | Medical History | 25 |
| <i>8.6.2</i> . | · | |
| 8.6.2 | 2.1. Extent of Exposure | 25 |
| 8.6.2 | 1 | |
| 8.6.3. | Adverse Events | |
| 8.6.4. | Clinical Laboratory Evaluations | |
| 8.6.5. | Vital Signs | |
| 8.6.6. | Physical Examination | |
| 8.6.7. | ECG | |
| 8.6.8. | Subjective Opiate Withdrawal Scale (SOWS) | |
| 8.6.9.<br><b>8.7</b> | Pharmacokinetic Procedures | |
| 8.7.1. | | |
| 8.7.2. | | |
| | 1 | |
| | MPUTER SOFTWARE | |
| 10. RE | FERENCES | 29 |
| 11. AP | PENDICES | 29 |
| 11.1 | APPENDIX 1: VARIABLE DEFINITIONS | 29 |

Client: Trevena, Inc. Protocol/CIP #: CP130-3003

Version #: 1.0


## 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# **Table 1: Abbreviations and Definitions of Terms**

| ACEP | American College of Emergency Physicians |
|--------|------------------------------------------------|
| AEs | adverse events |
| ALT | alanine aminotransferase |
| AST | Asparate aminotransferase |
| ASA | American Society of Anesthesiologists |
| bmi | body mass index |
| BP | blood pressure |
| bpm | beats per minute |
| cm | centimeters |
| °C | Celsius |
| CRF | case report form |
| CYP | cytochrome P450 enzyme (e.g. CYP2D6) |
| DBP | diastolic blood pressure |
| DOB | date of birth |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EDs | emergency departments |
| ESI | Emergency Severity Index |
| FDA | Food and Drug Administration |
| °F | Fahrenheit |
| HR | heart rate |
| ICD | International Classification of Diseases |
| ICF | informed consent form |
| IP | investigational product |
| IV | intravenous |
| kg | Kilograms |
| max | Maximum |
| MedDRA | medical dictionary for regulatory activities |
| mg | Milligram |
| min | Minimum |
| MRPSS | Moline-Roberts Pharmacologic Sedation Scale |
| NPRS | numeric pain rating scale |
| PACU | post-anesthesia care unit |
| PCA | patient-controlled analgesia device |
| PCSA | Potentially Clinically Significant Abnormality |
| PK | pharmacokinetic |
| PRN | as needed |
| PT | preferred term |
| 1.1 | profession term |


Protocol/CIP#: CP130-3003

| QT <sub>c</sub> | Q-T interval corrected for heart rate |
|---|---|
| $QT_{c}F$ | Q-T interval corrected for heart rate using Frederica's formula |
| RR | respiration rate |
| SAEs | erious adverse events |
| $SAS^{(\! R \! \!$ | statistical analysis software |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SOC | system organ class |
| SOP | standard operating procedures |
| SOWS | Subjective Opiate Withdrawal Scale |
| TEAE | treatment-emergent adverse event |
| TEMP | Temperature |
| $t_x$ | Time from the start of dose $(t_0)$ |
| WHO | World Health Organization |

### 2. INTRODUCTION

Inadequately treated pain has significant short- and long-term consequences, including prolonged emergency stays, psychological disturbances, and dissatisfaction with medical care. Opioid analgesics like morphine, fentanyl, and hydromorphone are mainstays of acute pain management; however, their use is hampered by well-known adverse events (AEs), such as respiratory depression, nausea, vomiting, and sedation (Lubawski, 2008) (Philip, 2002). Ultimately, the unmet medical need in acute pain therapy is an increased level of efficacy with acceptable tolerability.

This is a phase III, multicenter, open-label study to evaluate the safety of oliceridine (TRV130) in patients with moderate to severe acute pain for which parenteral opioid therapy is warranted.

This study will be conducted in inpatient hospitals, outpatient hospital departments, ambulatory surgical care centers, and emergency departments (EDs). Patients recruited in EDs may continue oliceridine treatment if hospitalized and parenteral opioid therapy is warranted.

Representative surgeries include orthopedic, abdominal, gynecological, vascular, soft tissue, and surgical procedural pain.

Representative medical conditions include acute pancreatitis, acute exacerbation of existing noncancerous chronic pain, musculoskeletal pain, sickle-cell disease, inflammatory orofacial muscle pain, and renal colic. Medical conditions that could confound the evaluation of oliceridine are excluded, such as acute pain without a specific etiology, undifferentiated acute abdominal pain, acute breakthrough pain in palliative "end of life" care, and pain associated with advanced cancer (somatic, visceral, or neuropathic) or with concurrent use of chemotherapeutic or biologic agents for the treatment of cancer.


Protocol/CIP#: CP130-3003

Representative ED conditions include visceral pain (eg, renal colic, upper abdominal pain, abdominal pelvic pain); nonvisceral pain (eg, traumatic and atraumatic acute musculoskeletal pain, chest wall pain, burns, orofacial pain/headache, cutaneous and soft tissue pain); procedural analgesia (eg, reduction of orthopedic fractures and dislocations, abscess incision and drainage); acute painful episodes associated with a medical condition (eg, sickle cell painful vaso-occlusive episode). Oliceridine will not be used to intentionally suppress a patient's level of consciousness (procedural sedation and analgesia as defined by the American College of Emergency Physicians [ACEP]).

### 3. STUDY OBJECTIVES

The primary objective is to evaluate the safety and tolerability of oliceridine in patients with moderate to severe acute pain for which parenteral opiod therapy is warranted.

The secondary objective is to evaluate the analgesic efficacy of oliceridine.

### 4. STUDY DESIGN

#### 4.1 General Design

This is a phase III, multicenter, open-label study to be conducted in four phases: Screening/Baseline, Treatment (consisting of a pre-dose period and a dosing period), End-of-Treatment, and Follow-up.

During the screening phase, patients will provide written informed consent before any protocol-specified procedures or assessments are performed. All screening procedures will be completed within 14 days before the first oliceridine dose. Select standard of care assessments (e.g., chemistry, hematology, urine or serum pregnancy test, urine or serum toxicology screen, electrocardiogram (ECG)) obtained before informed consent may be used as study data if protocol specifications and timeframes are met (see Protocol Section 3.6.1). When screening and baseline procedures are anticipated to occur within 48 hours of each other, they may be executed as a single procedure, unless the clinical condition of the patient has significantly changed since screening.

The treatment phase begins with the pre-dose period and ends when the investigator documents that the last dose of oliceridine was administered and that the patient will no longer be treated with oliceridine. The duration of treatment for each patient will be determined by the clinical need for parenteral opioid therapy. In current practice, parenteral opioids are used as-needed for up to several days. Although preclinical toxicology studies support intravenous (IV) administration of oliceridine for up to 14 days, it is unlikely that patients will receive oliceridine for that duration in the context of this study.

Before dosing with oliceridine, vital signs, oxygen saturation, and somnolence/sedation will be measured. Pre-dose period procedures will occur within 30 minutes before the first oliceridine dose and if the dosing period is delayed, pre-dose period procedures will be repeated. An


Protocol/CIP#: CP130-3003

additional post-surgical ECG will be performed only in surgical patients. Prior medications and AEs/SAEs will be recorded. Pain intensity will be measured using a 0-10 point numeric pain rating scale (NPRS).

Oliceridine IV infusion may be administered either by clinician-administered bolus, patient-controlled analgesia device (PCA), or both bolus and PCA, according to the clinical situation. During dosing with oliceridine, vital signs, oxygen saturation, and somnolence/sedation will be measured at any and all times during the dosing period consistent with individual patient need and institutional standards of care for a patient receiving a parenteral opioid. An ECG will be obtained 60 minutes after the first dose of oliceridine, and at every 24 hours of oliceridine treatment. Blood will be collected for clinical laboratory tests, oliceridine pharmacokinetics and future cytochrome P450 2D6 (CYP2D6) genotyping. Concomitant medications and AEs/SAEs will be recorded. NPRS assessment will also be completed at 30 minutes +/-10 minutes after the first dose of oliceridine and at any and all times during the dosing period consistent with individual patient need and institutional standards of care for a patient receiving a parenteral opioid.

When the investigator documents that the last dose of oliceridine was administered and that the patient will no longer be treated with oliceridine, the treatment phase is complete and the end-of-treatment phase begins. A physical examination will be performed at this time. Within 1 hour after completion of the treatment phase, vital signs, oxygen saturation, and somnolence/sedation will be measured, and concomitant medications and AEs/SAEs will be recorded. Within 3 hours after completion of the treatment phase, blood will be collected for clinical laboratory tests. Concomitant medications and AEs/SAEs will be recorded. Patients will be observed for at least 3 hours after the last dose of oliceridine; however, medically-required transfer of an ED patient to another facility takes precedence over study procedures. The Subjective Opioid Withdrawal Scale (SOWS) will be administered to detect symptoms of opioid withdrawal. If the patient is discharged or transferred before the time when the SOWS is to be performed, it will be performed 1 day after completion of the treatment phase and returned to the site by mail or in person.

A follow-up contact will be made between 2 and 3 days after completion of the treatment phase. The contact may be conducted in person or by telephone. Concomitant medications and AEs/SAEs will be recorded. The surgical procedure, medical diagnosis or ED diagnosis for which parenteral opioid therapy was warranted will be captured using the International Classification of Diseases, 10<sup>th</sup> Revision (ICD-10) terminology.

A flow chart of the study design is presented below:


Protocol/CIP #: CP130-3003



Abbreviations:  $t_0$  = time of first dose of oliceridine; h = hours

## 4.2 Method of Assignment of Patients to Cumulative Dose Groups

This is an open-label study therefore the method of assigning patients to dose groups will be based on the actual dose received by the patient.

Depending on the clinical considerations for which parenteral opioid therapy is warranted (e.g., anticipated duration of therapy, clinical site/setting), a patient could receive oliceridine using clinician-administered bolus dosing or PCA dosing. For clinician-administered bolus dosing, the oliceridine initial dose is 1 mg to 2 mg. If clinically indicated, a 1 mg supplemental dose may be administered as early as 15 minutes after the initial dose. Subsequent doses are 1 to 3 mg every 1 to 3 hours PRN based on individual patient need and previous response to oliceridine. In settings where rapid analgesia is targeted (e.g., ED or post-anesthesia care unit (PACU)), the oliceridine initial dose is 1 mg to 3 mg. If clinically indicated, 1 mg to 3 mg supplemental doses may be administered every 5 minutes PRN. Subsequent doses are 1 to 3 mg every 1 to 3 hours PRN based on individual patient need and previous response to oliceridine. For PCA dosing, the oliceridine regimen will consist of a loading dose, a demand dose, and a lockout interval without a continuous baseline infusion.

## Oliceridine PCA regimen:

- Loading dose: 1.5 mg.
- Demand dose: 0.5 mg.
- Lockout interval: 6 minutes.

If clinically indicated, throughout the treatment phase, a 1 mg supplemental dose may be administered PRN, taking into account the patient's utilization of PCA demand doses, individual patient need and previous response to oliceridine.

For purposes of analysis the cumulative dose groups will be grouped in the following categories where cumulative dose group will be defined as the sum of all individual doses:

<sup>\*</sup> Combined if occurring within 48 hours of each other, unless the clinical condition of the patient has significantly changed since screening.

Client: Trevena, Inc. Protocol/CIP #: CP130-3003


Oliceridine Oliceridine Oliceridine Oliceridine Oliceridine All Treated <= 4 mg >4 to 8 mg >8 to 16 mg >16 to 36 mg >36 mg Patients

## 4.3 Blinding

This is an open-label trial in which all patients will receive oliceridine; therefore, blinding is not applicable.

## 4.4 Determination of Sample Size

No formal sample size calculations were made. Approximately 1000 patients will be treated with oliceridine.

#### 5. CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

At the time of the writing of this document, protocol amendment 5 has been approved. For changes in the conduct of the study or planned analyses, please see the individual protocol amendments.


Protocol/CIP #: CP130-3003

PCN #: 2jk00017

## 6. BASELINE, SAFETY & TOLERABILITY, EFFICACY and PHARMACOKINETIC EVALUATIONS

#### **6.1** Schedule of Evaluations

| | Screening<br>phase <sup>1</sup> | | | ent phase<br>14 days) | End | -of-treatment p | ohase <sup>2</sup> | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedures | (<= 14<br>days<br>before<br>first dose<br>of<br>oliceridin<br>e) | Baselin<br>e<br>phase <sup>1</sup><br>(Day 1) | Predose<br>(Day 1) | T0 to last<br>dose of<br>oliceridine | End-of-<br>treatment<br>documentati<br>on <sup>2</sup> | Within<br>1hour after<br>completion<br>of treatment<br>phase <sup>2</sup> | Within<br>3 hours after<br>completion of<br>treatment<br>phase <sup>2</sup> | One day<br>after<br>completion<br>of treatment<br>phase | Follow-up phase <sup>3</sup> (Between 2 days and 3 days after completion of treatment phase) |
| Informed consent <sup>5</sup> | X | | | | | | | 1000 | 200 |
| Demographics | X | | | | | | | | |
| Medical history | X | X | | | | | | | |
| Eligibility criteria | X | X | | | | | | | |
| ASA physical status<br>classification <sup>6</sup> | X | X | | | | | | | |
| ESI <sup>7</sup> | X | | | | | | | | |
| Physical examination <sup>2</sup> | X | X | | | X | | | | |
| Clinical laboratories8 | X | X | | | | | X | | |
| Blood sample for future<br>CYP2D6 genotyping | | | | X | | | | | |
| Urine or serum<br>pregnancy test <sup>9</sup> | X | X | | | | | | | |
| Urine or serum<br>toxicology screen <sup>10</sup> | X | | | | | | | | |
| Weight | X | X | | | | | | | |
| Height <sup>11</sup> | X | | | | | | | | |
| ECG | X | X | $X^{12}$ | $X^{13}$ | | | | | |
| PK sampling <sup>14</sup> | | | | X | | | | | |
| PCA patient training <sup>15</sup> | X | X | X | X | | | | | |
| Oliceridine dosing | | 200.00 | .0110000 | X | | | | | |
| NPRS <sup>16</sup> | | X | X | X | | X | | | |
| Vital signs <sup>17</sup> | X | X | X | X | | X | | | |
| MRPSS <sup>18</sup> | | | X | X | | X | | | |
| SOWS <sup>19</sup> | | | | | | | | X | |
| Oxygen saturation <sup>20</sup> | | | <b>←</b> | <b>Υ</b> | | | | | |
| Prior, concomitant<br>medications <sup>21</sup> | <b>←</b> | X | <del>-</del> | ← | | | X | | ······································ |
| AE/SAE reporting <sup>22</sup> | <b>←</b> | | | | | X | | | → |

Abbreviations: AE = adverse event; ASA = American Society of Anesthesiologists; CYP2D6 = cytochrome P450 2D6; ECG = electrocardiogram; ESI = Emergency Severity Index; MRPSS = Moline-Roberts Pharmacologic Sedation Scale; NPRS = Numeric Pain Rating Scale; PCA = patient-controlled analgesia device; PK = pharmacokinetic; SAE = serious adverse event; SOWS = Subjective Opiate Withdrawal Scale; T0 = time of first oliceridine dose.

Chiltern, International – Confidential

Chiltern, International, All rights reserved. Reproduction or transmission to others apart from the parties involved with this document in any form or by any means is not permitted without the prior written consent of Chiltern, International.


Protocol/CIP #: CP130-3003

PCN #: 2jk00017

- 1. When screening and baseline procedures are anticipated to occur within 48 hours of each other, they may be executed as a single procedure, unless the clinical condition of the patient has significantly changed since screening.
- 2. When the investigator documents that the last dose of oliceridine was administered and that the patient will no longer be treated with oliceridine, the treatment phase is complete and the end-of-treatment phase begins. A physical examination will be performed at this time.
- 3. Follow-up contact may be conducted in person or by telephone.
- 4. Procedures will be performed at any and all times during the dosing period consistent with individual patient need and institutional standards of care for a patient receiving a parenteral opioid.
- 5. Written informed consent.
- 6. If a surgical or medical patient. Refer to Section 9.3 of the protocol for the ASA scale.
- 7. If an ED patient. Refer to Section 9.4 of the protocol for the ESI scale.
- 8. Blood chemistry and hematology will be obtained using local laboratories and local laboratory range values.
- 9. Female patients of childbearing potential only.
- 10. If an ED patient.
- 11. Height may be obtained by measurement or patient attestation.
- 12. During the pre-dose period, an additional, post-surgical ECG will be performed only in surgical patients.
- 13. ECG will be obtained during the Treatment Phase at 60 minutes after the first dose of oliceridine, and at every 24 hours of oliceridine treatment.
- 14. PK samples will be collected at two times during the treatment phase: sample 1 at 30 minutes (+/- 10 minutes) after the first dose; sample 2 between 1 and 2 hours after the first dose. Unscheduled PK samples may be required. Refer to Sections 3.5.2.3 and 3.6.3 of the protocol.
- 15. PCA patient training is required before PCA use. If PCA is planned, training will occur during the screening and baseline phases; if PCA is started during the treatment phase, training will occur before PCA use. Training is repeated according to patient need.
- 16. NPRS will be measured during the pre-dose period, at 30 minutes +/-10 minutes after the first dose of oliceridine, and at any and all times during the dosing period consistent with individual patient need and institutional standards of care for a patient receiving a parenteral opioid (see Section 9.2 of the protocol).
- 17. Blood pressure, heart rate, respiratory rate, and temperature. Temperature will be measured at screening and baseline only.
- 18. Refer to Section 9.1 of the protocol for the MPRSS.
- 19. Refer to Section 9.5 of the protocol for the SOWS. If the patient is discharged or transferred before the time when the SOWS is to be performed, it will be performed one day after completion of the treatment phase and returned to the site by mail or in person.
- 20. Oxygen saturation monitoring will be continuous but will be recorded at any and all times during the dosing period consistent with individual patient need and institutional standards of care for a patient receiving a parenteral opioid. The date and time of initiation and discontinuation of continuous oxygen saturation monitoring will be recorded in the source documents.
- 21. Prior medications are defined as those taken before the first dose of oliceridine. Concomitant medications are defined as those taken after the first dose of oliceridine. Prior medications taken or administered within the 14 days before the first dose of oliceridine will be recorded in source and will also be recorded in eCRF. Supplemental oxygen will be recorded as a prior and/or concomitant medication.
- 22. AEs occurring from time of informed consent to the follow-up phase will be recorded in source and will also be recorded in eCRF if the patient receives oliceridine. SAEs occurring from time of informed consent to the follow-up phase or 7 days after the last dose of oliceridine (whichever occurs later) will be recorded in source and eCRF; ongoing SAEs after this time frame will be followed until the investigator, medical monitor, and sponsor agree that the SAE is satisfactorily resolved. SAEs considered by the investigator to be related to oliceridine, regardless of the time of onset after treatment, should be reported.


Protocol/CIP #: CP130-3003 Client: Trevena, Inc.


### **6.2** Time Point Algorithms

#### **6.2.1.** Baseline Assessments

Baseline assessments are listed in Section 3.6.1 of the study protocol. In general, baseline values will be defined as the last non-missing value (scheduled, unscheduled or repeat) prior to the patient receiving the first dose of oliceridine.

The following assessments will have a baseline value:

- **NPRS**
- Clinical Laboratories
- Vital Signs
- MRPSS Total Score
- ECG

## 6.2.2. Initial Setting and Condition Category

During the screening phase, the initial setting (Surgical, Medical and ED) will be recorded. The condition category for which parenteral opioid therapy was warranted will be captured using the International Classification of Diseases, 10<sup>th</sup> Revision (ICD-10) terminology.

#### **6.2.3.**Relative Day

The date of the first dose of oliceridine will be considered relative day 1, and the day before the first dose of oliceridine will be relative day -1. Relative days for events on or after the first dose will be calculated as date of event - date of first dose of oliceridine + 1. Relative days for events before the first dose will be calculated as date of event - date of first dose of oliceridine.

Study hour will be calculated relative to the first dose of oliceridine also: date/time of event - date/time of first dose of study drug.

#### **6.2.4.** Analysis Windows

All NPRS, PK, ECG, Cumulative Exposure, Laboratory Assessments, Vital Signs, Oxygen Saturation, and MRPSS data collected during the treatment period will be windowed to an appropriate analysis time window based on the following time intervals.

# Analysis Windows for Exposure, Laboratory Assessments,

| Vit | al Signs, Oxygen Saturation, a | and MRPSS |
|-----|--------------------------------|-----------|
| nt | Analysis Window | Midpoin |

| Windowed Time Point | Analysis Window | Midpoint of Analysis Window |
|---------------------|------------------------|-----------------------------|
| Baseline | <0 minutes | NA |
| T30 minutes | $\geq 0 - \leq 1$ hour | 30 minutes |
| T2.5 hours | ≥1 -<4 hours | 2 hours and 30 minutes |
| T8 hours | $\geq$ 4 – <12 hours | 8 hours |
| T18 hours | ≥12 – <24 hours | 18 hours |


Client: Trevena, Inc. Protocol/CIP #: CP130-3003


| T30 hours | ≥24 – <36 hours | 30 hours |
|-----------|-----------------|----------|
| T42 hours | ≥36 – <48 hours | 42 hours |
| T60 hours | ≥48 – <72 hours | 60 hours |
| T84 hours | ≥72 – <96 hours | 84 hours |
| T96 hours | ≥96 hours | 96 hours |

## **Analysis Windows for ECG**

| <b>Windowed Time Point</b> | Analysis Window | Midpoint of Analysis Window |
|---|---|---|
| Baseline | <0 minutes | NA |
| T60 minutes | $\geq 0 - < 1.5 \text{ hours}$ | 1 hour |
| T6 hours | $\geq 1.5 - < 12 \text{ hours}$ | 6 hours |
| T24 hours | $\geq$ 12 – <36 hours | 24 hours |
| T48 hours | $\geq$ 36 – <63 hours | 48 hours |
| T72 hours | ≥63 – <96 hours | 72 hours |
| T96 hours | ≥96 hours | 96 hours |

#### **Analysis Windows for NPRS**

| Windowed Time Point | Analysis Window | Midpoint of Analysis Window |
|---|---|---|
| Baseline | <0 minutes | NA |
| T20 minutes | ≥0 - <40 minutes | 30 minutes |
| T1 hour | $\geq$ 40 – <1.5 hour | 1 hour |
| T3.5 hours | $\geq 1.5 - < 6$ hours | 3 hours and 45 minutes |
| T12 hours | $\geq 6 - \leq 14 \text{ hours}$ | 10 hours |
| T19 hours | ≥14 – <24 hours | 19 hours |
| T24 hours | ≥24 hours | 24 hours |

## **Analysis Windows for PK**

| <b>Windowed Time Point</b> | Analysis Window | <b>Protocol Allowed Window</b> |
|---|---|---|
| Baseline | ≤0 minutes | NA |
| T30 minutes | >0 – <1 hour | ±10 minutes |
| T1.5 hours | $\geq 1 - \leq 2$ hours | $\geq 1 - \leq 2$ hours |
| T14 hours | $\geq$ 2 – <24 hours | NA |
| T36 hours | ≥24 – <48 hours | NA |
| T60 hours | ≥48 – <72 hours | NA |
| T84 hours | ≥72 –<96 hours | NA |

Unless stated otherwise, if multiple observations fall within the same analysis window, the measurement closest to the midpoint of the analysis time point will be selected. If there are more than 1 assessments equal distant from the midpoint of the analysis time point, the later of the data points will be used in the analysis. All selected observations will be flagged in the listings and only the flagged observation will be used in the descriptive summary statistics over time for each parameter.

Client: Trevena, Inc. Protocol/CIP #: CP130-3003


In addition to the windowed values collected during the treatment phase, the protocol specified assessments for vital signs, oxygen saturation, MRPSS and laboratory End-of-Treatment values will be summarized using descriptive statistics. The End-of-Treatment values are defined as the first observation after the end of study date/time.

### **6.3** Safety Assessments

### 6.3.1 Extent of Exposure

Depending on the clinical considerations for which parenteral opioid therapy is warranted, a patient could receive oliceridine using clinician-administered bolus dosing or PCA dosing. Patients will have the method of administration categorized as PCA if they received at least 1 PCA dosing. Otherwise the method of administration will be categorized as bolus.

Duration is defined as the difference in total hours from the first dose to the last dose of study medication.

### 6.3.2 Adverse Events

Adverse events includes any newly occurring event or previous condition that increased in severity or frequency from time of informed consent. AEs occurring from time of informed consent to the follow-up phase will be recorded in source documentation and will also be recorded in the EDC system if the patient receives oliceridine. All AEs must be recorded irrespective of whether or not they are considered medication-related. All AEs that are possibly or probably related to study medication will be followed until resolution or database lock, whichever occurs first. Changes in intensity or frequency of AEs should be recorded as separate events (i.e., a new record started).

Treatment emergent adverse events (TEAEs) are defined as AEs with onset at the time of or following the start of treatment with study medication until 7 days after the last dose of study medication or any pre-existing AEs that have worsened in severity on or after the first dose of study medication and through 7 days after the last dose of study medication.

Adverse events will be designated as treatment-emergent according to the following algorithm:

- If both the start date and start time of an AE are known, then:
- If the AE starts at any time prior to the time of the first dose on Day 1, then the AE will not be designated as treatment-emergent and hence will not be summarized.
- If the AE starts on or after the time of the first dose on Day 1 through 7 days after the last dose, then the AE will be designated as treatment-emergent.
- If only the start date of an AE is known and the start time of the AE is unknown, then:
- If the AE starts on Day 0, then the AE will not be designated as treatmentemergent and hence will not be summarized.

Protocol/CIP#: CP130-3003 Client: Trevena, Inc.


• If the AE starts on Days 1 through 7 days after the last dose, then then the AE will be designated as treatment-emergent.

All AEs will be assessed on two descriptive parameters: intensity and relationship to the study medication:

• Intensity refers to the severity of an event and references impact on a patient's functioning. The following categories will be used to classify intensity:

Mild Awareness of sign or symptom, but easily tolerated

Moderate Discomfort enough to cause interference with usual activity

Severe Incapacitating with inability to work or perform usual activity

• Relationship refers to the likelihood that the event being assessed was caused by the study medication. The following categories will be used to classify relationship:

**Not Related** There is no reasonable association between the study

treatment and the suspected event.

Unlikely It is doubtful that there is an association between the study

treatment and the suspected event. The event could have Related

been produced by the patient's clinical state or other modes

of therapy administered to the patient.

**Possibly** The suspected AE may or may not follow a reasonable Related

temporal sequence from study treatment administration. The

event could have been produced or mimicked by the patient's clinical state or by other modes of therapy

concomitantly administered to the patient.

**Probably** The suspected AE follows a reasonable temporal sequence

from study treatment administration, abates upon Related

> discontinuation of the treatment, and cannot be reasonably explained by the known characteristics of the patient's

clinical state.

For summaries by relationship, possibly and probably related will also be combined into one "related" summary.


#### 6.3.3 Clinical Laboratory Evaluations

Baseline values are defined as the last measurements taken before the first dose of oliceridine. Change from baseline will be defined as the post baseline value minus the baseline value.

The investigator will exercise his or her medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.

Liver chemistry thresholds have been designed to assure patient safety. When patients meet the hepatic transaminase threshold criteria (AST or ALT >=3 × upper limit of normal [ULN]), the patient should undergo close observation, including monitoring for symptoms (clinical symptoms of hepatitis or hypersensitivity, fatigue, decreased appetite, nausea, vomiting, abdominal pain, jaundice, fever, or rash) and hepatic function (AST, ALT, alkaline phosphatase, and fractionated bilirubin) at least every 48 hours, until symptoms and/or hepatic function abnormalities resolve, stabilize, or return to baseline values. The following thresholds will be derived and presented for hepatic chemistry:

- AST  $\geq$  3 x ULN
- ALT  $> 3 \times ULN$
- AST or ALT  $\geq$  3 x ULN
- AST  $\geq$  5 x ULN
- ALT  $\geq$  5 x ULN
- AST or ALT  $\geq$  5 x ULN
- BILI  $\geq 2 \times ULN$

## 6.3.4 Vital Signs

Baseline values are defined as the last measurements taken before the first dose of oliceridine. Change from baseline will be defined as the post baseline value minus the baseline value. Vital signs will include blood pressure (BP), heart rate (HR), respiratory rate (RR), and temperature. Temperature will be measured at screening and baseline only.

Potentially clinically significant abnormal (PCSA) vital signs parameter criteria is defined below:

| Parameter | Criterion value | Change relative to baseline |
|---|---|---|
| Systolic blood pressure (mmHg) | $\geq$ 180 mmHg | 25% increase |
| Systolic blood pressure (mmHg) | $\leq 80 \text{ mmHg}$ | 25% decrease |
| Diastolic blood pressure (mmHg) | ≥ 110 mmHg | 25% increase |
| Diastolic blood pressure (mmHg) | $\leq$ 40 mmHg | 25% decrease |
| Pulse rate (bpm) | ≥ 120 bpm | 15 bpm increase |
| Pulse rate (bpm) | ≤ 40 bpm | 15 bpm decrease |


#### 6.3.5 Electrocardiogram (ECG)

ECG summaries will include HR, PR interval, RR interval, QRS interval, QT interval, and QTcF interval. Baseline values are defined as the last measurements taken before the first dose of oliceridine. Change from baseline will be defined as the post baseline value minus the baseline value.

In addition to the observed values for these parameters, the following will be categorized:

- Change from Baseline QTcF > 30 milliseconds
- Change from Baseline QTcF > 60 milliseconds
- Increase of QTcF to > 500 milliseconds

The investigator will exercise his or her medical and scientific judgment in deciding whether an abnormal finding is clinically significant.

## 6.3.6 Physical Examination

The physical examination will include general appearance. Results from screening/baseline will be recorded as medical history events while changes from screening/baseline in the physical examination will be recorded as AEs. The investigator will exercise his or her medical and scientific judgment in deciding whether an abnormal finding is clinically significant.

#### 6.3.7 Subjective Opiate Withdrawal Scale (SOWS)

The Subjective Opioid Withdrawal Scale (SOWS) will be administered one day after completion of the treatment phase to detect symptoms of opioid withdrawal. Patients will score each of the 16 symptoms on an intensity scale ranging from 0 "not at all" to 4 "extremely".

If the patient is discharged or transferred before the time when the SOWS is to be performed, it will be performed one day after completion of the treatment phase and returned to the site by mail or in person.

Each patient should have exactly one SOWS administered during the study. However, if multiple SOWS results are collected for any given patent, the record with the most extreme total score will be used for summary purposes.

### 6.3.8 Oxygen Saturation

Baseline values are defined as the last measurements taken before the first dose of oliceridine. Change from baseline will be defined as the post baseline value minus the baseline value.

Potentially clinically significant abnormal (PCSA) oxygen saturation criteria is defined below:

Client: Trevena, Inc. Protocol/CIP #: CP130-3003


| Parameter | Criterion value | Change relative to baseline |
|-------------------|-----------------|-----------------------------|
| Oxygen Saturation | < 90 % | NA |

## 6.3.9 Somnolence/Sedation

The Moline-Roberts Pharmacologic Sedation Scale (MRPSS) will be used to measure somnolence/sedation. Baseline values are defined as the last measurements taken before the first dose of oliceridine. Six levels describe the range of sedation from "none to minimal" to "general anesthesia":

| Presentation | Auditory<br>Stimulus | Tactile<br>Stimulus | Response | Sedation |
|---|---|---|---|---|
| Awake, aware, alert<br>Airway and ventilation<br>adequate | None | None | Spontaneous,<br>sustained<br>interaction | 1<br>None to Minimal |
| Restful, drowsy, dozing,<br>lightly sleeping<br>Airway and ventilation<br>adequate | Soft voice or ambient noise | None or light touch, rubbing or tapping | Sustains<br>interaction | 2<br>Anxiolysis |
| Sleeping<br>Airway and ventilation<br>adequate | Soft to normal voice | Light touch,<br>rubbing or<br>tapping | Limited or brief interaction | 3<br>Moderate<br>Sedation |
| Sleeping<br>Airway and ventilation<br>adequate | Normal to loud voice | Light touch,<br>rubbing or<br>tapping | Follows simple commands | 4<br>Moderate<br>Sedation |
| Sleeping<br>Airway and ventilation<br>may be impaired | Loud voice | Intense to noxious | Purposeful<br>response or<br>non-purposeful | 5<br>Deep<br>Sedation |
| Sleeping<br>Airway and ventilation<br>likely impaired | Loud voice | Noxious | No response, unarousable | 6<br>General<br>Anesthesia |

#### **6.4** Drug Concentration Measurements and Pharmacokinetic Parameters

For all samples, the actual sampling time will be recorded.

## 6.5 Efficacy Variables

## 6.5.1. Numeric Pain Rating Scale (NPRS)

The NPRS is a generic, unidimensional questionnaire of pain intensity in adults. In the NPRS, a respondent selects a whole number (0-10 integers) on a single 11 point scale that best reflects the intensity of their pain. In this scale, the 0 is anchored with the descriptor "no pain" and the 10 is anchored with the descriptor "worst pain imaginable". Baseline values are defined as the last measurements taken before the first dose of oliceridine. Change from baseline will be defined as the post baseline value minus the baseline value.


#### 7. STATISTICAL METHODS

## 7.1 General Methodology

Data will be summarized using descriptive statistics (number of patients [N], mean, standard deviation [SD], median, minimum, and maximum) for continuous variables and using frequency and percentage for discrete variables. Unless specified otherwise, all summaries will be performed using SAS® Version 9.3 or higher.

## 7.2 Adjustments for Covariates

Not applicable to this study.

## 7.3 Handling of Dropouts or Missing Data

All dates presented in the individual patient listings will be as recorded on the eCRF, not as per the rules below. All rules explained below for partial/missing dates will be followed unless contradicted by any other data recorded on the electronic Case Report Form (eCRF).

#### 7.3.1. Adverse Events

If the AE stop date is completely missing and the AE has resolved, the stop date will be imputed as the date of the patient's last visit in the study.

- If only the year is known, the stop date will be imputed as "31-Dec" of that year or as the date of the patient's last clinic visit in the study if in the same year.
- If the month and year are known, the stop date will be imputed as the last day of that month unless the stop date corresponds to the same month as the patient's last clinic visit in which case the date of patient's last clinic visit in the study will be used instead.

If the start date is completely missing it will be imputed as follows:

- If the stop date occurs on or after the start of study medication or the event is
  ongoing, the start date will be imputed as the date of the first dose of study
  medication.
- If the stop date occurs before the start of study medication, the start date of the event will be imputed as the patient's screening date or the stop date of the event, whichever the earlier.

If the start time is missing it will be imputed only in the case where the start date of the event corresponds to the date of the first dose of study medication. In this case the time will be imputed as the same time as the first dose of study medication. In all other cases the time will not be imputed. Imputed dates will be used for calculations, however the actual date collected will be presented in listings.


### 7.3.2. Concomitant Medications

If the stop date is completely missing and the patient has stopped taking the CM, the stop date will be imputed as the date of the patient's last visit in the study.

- If only the year is known, the stop date will be imputed as "31-Dec" of that year or as the date of the patient's last clinic visit in the study if in the same year.
- If the month and year are known, the stop date will be imputed as the last day of that month unless the stop date corresponds to the same month as the patient's last clinic visit in which case the date of patient's last clinic visit in the study will be used instead.

If the start date is completely missing it will be imputed as follows:

- If the stop date occurs on or after the start of study medication or the concomitant medication is ongoing, the start date will be imputed as the date of the first dose of study medication.
- If the stop date occurs before the start of study medication, the start date of the medication will be imputed as the patient's screening date or the stop date of the medication whichever the earlier.

If the start time is missing it will be imputed only in the case where the start date of the medication corresponds to the date of the first dose of study medication. The time will be imputed as the same time as the first dose of study medication. In all other cases the time will not be imputed. Imputed dates will be used for calculations, however the actual date collected will be presented in listings.

## 7.3.3. Study Medication Dosing

The start date/time of first dose of study medication is not expected to be missing for any patient in the Safety Analysis Set. If the stop date/time of last dose of study medication is completely missing, then the date/time of last dose of study medication will be assigned as the earliest of the 5 options below for analysis purposes:

- 1. Start date/time of last dose
- 2. Date/time from end of treatment phase declaration
- 3. Date/time of patient's first end-of-treatment phase assessment in the study
- 4. Early termination
- 5. Death (assuming time of death of 23:59 if only date is available; time may be obtained from stop time of associated AE with fatal outcome)

Client: Trevena, Inc. Protocol/CIP #: CP130-3003


## 7.3.4. Medical History

If the month and year are present but the day is missing, the diagnosis date will be set to first day of the relevant month. If only the year is recorded, the diagnosis date will be set as "01-Jan" for that year. If the entire date is missing, the start date of diagnosis will remain missing.

## 7.3.5. Numeric Pain Rating Scale

For patients who have no NPRS assessments recorded prior to the first dose of study medication, the baseline will be imputed with a score of 4. Otherwise, there will be no imputation of missing data for NPRS.

## 7.3.6. Subjective Opioid Withdrawal Scale

Opioid withdrawal will be measured using the Subjective Opioid Withdrawal Scale (SOWS) consisting of 16 symptoms rated in intensity (0=Not at all, 1=A little, 2=Moderately, 3=Quite a bit, 4=Extremely). The total score will be derived by summing the individual symptom intensities and will range from 0 to 64. If there are no more than half of the symptoms that are missing from the SOWS, imputation with the mean score of the non-missing questions will be used to calculate total score. SOWS with more than half of the symptoms missing will have total score missing.

### 7.4 Interim Analyses and Data Monitoring

No data monitoring committees are planning for this study. An interim analysis is expected to be performed in order to support regulatory discussions. No statistical testing will be performed.

## 7.5 Multi-Center Studies and Pooling of Centers

This study will be conducted at approximately 60-90 study centers located in the United States. No pooling of the sites will be performed since no formal statistical tests will be performed for the different centers.

## 7.6 Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons or multiplicity will be made.

## 7.7 Examination of Subgroups

The analysis of safety will be examined by looking at the following subgroups: sex (females vs. males); age grouping 1 (<65 years vs. ≥65 years); age grouping 2 (≥18 to <study median years of safety analysis set population vs. ≥study median years of safety analysis set population); race (white vs non-white); median baseline NPRS score (< median vs. ≥ median); initial setting, BMI (<25 vs. >=25), and CYP2D6 metabolizer status.

No statistical testing will be performed for the subgroup analyses but any differences in treatment effect noticed in subgroups may be explored.


Client: Trevena, Inc. Protocol/CIP #: CP130-3003


### 8. STATISTICAL ANALYSIS

The standard operating procedures (SOPs) of Chiltern, International, will be followed in the creation and quality control of all data displays and analyses.

## 8.1 Disposition of Subjects

The number of patients in each analysis set will be tabulated for all the Enrolled Analysis Set. Safety Analysis Set will be further summarized by each site and by cumulative dose group and all groups combined.

In addition, summary of reasons for screen failure will be tabulated for the Enrolled Analysis Set. The inclusion and exclusion criteria will be summarized in two separate categories. The inclusion criteria will be further categorized to patients not meeting the NPRS threshold and those not meeting other inclusion criteria. Patients with multiple reasons for failure or termination will be counted in each reason category.

Safety Analysis Set will be further summarized by cumulative dose group and all groups combined. The number of patients that completed the study, the number of patients that discontinued early, the number of patients for each reason for ealy discontinuation and the number of patients discontinuing at each study window will be summarized. Study window will be defined as the date and time of termination minus the date and time of first dose of oliceridine. The time point intervals are defined in section 6.2.4

Because the duration of treatment for each patient in this study will be determined by the clinical need for parenteral opioid therapy, a patient will be considered to be a completer if no early termination reason (e.g., AE to discontinuation, lack of efficacy) is indicated.

A listing with each patient's first/last dose of oliceridine, date/time of end of treatment, date of study completion and a potential reason for early termination will be provided. An additional listing with each patient's inclusion/exclusion criteria that caused the patients to be screen failures will be provided.

#### **8.2** Protocol Deviations

Protocol deviations will be listed by patient and summarized in a table based on protocol deviation categories as collected by the Kestrel clinical trial management system. This summary will be based on the Enrolled Analysis Set. Deviation categories will include procedure window, inclusion/exclusion criteria, unapproved medication, visit window, missed procedure, informed consent, and incorrectly performed procedure. A categorization of major or minor for each deviation will be determined by Trevena and recorded in the Kestrel database, as well as included as part of the summary table.

Protocol deviations will be summarized by cumulative dose groups based on their cumulative dose received. Screening failures will not be included in this summary. The categories will be sorted by descending count of patients in the all treated patients column.


#### **8.3** Analysis Populations

## 8.3.1. Enrolled Analysis Set

The enrolled population will include all patients that signed the informed consent form irrespective of whether they received oliceridine or not.

## 8.3.2. Safety Analysis Set

The safety analysis population will include all enrolled patients receiving at least 1 dose of oliceridine.

## 8.3.3. Efficacy Analysis Set

The efficacy analysis set will include all enrolled patients who received at least 1 dose of oliceridine and have at least 1 post-dose NPRS score.

## 8.4 Demographic and Other Baseline Characteristics

Demographic and baseline characteristics including age, height, weight, BMI, and baseline pain intensity will be summarized for each cumulative dose group and for all groups combined for the Safety Analysis Set with descriptive statistics (number of patients [n], mean, standard deviation [SD], median, minimum [min], and maximum [max]). No statistical comparisons will be performed for demographic and baseline characteristics.

Initial setting, gender, age groupings 1 and 2, race, race group, ethnicity, CYP2D6 metabolizer status, and BMI group will be summarized for each cumulative dose group and for all groups combined for the Safety Analysis Set using counts and percentages.

Data listings including demographic and baseline characteristics will be produced.

#### 8.5 Prior and Concomitant Medications

Prior and concomitant medications will be summarized separately using the Safety Analysis Set for each cumulative dose group and for all groups combined. The World Health Organization (WHO) Drug Dictionary, version March 2016, will be used to classify medications by preferred name and WHO ATC classification of ingredients. The number and percent of patients who took prior medications will be shown by WHO ATC classification of ingredients and by preferred term. The number and percent of patients who took concomitant medications will be shown in the same manner.

Data listings including prior and concomitant medications will be produced. Prior and concomitant medications will be distinguished directly in the listing.

#### 8.6 Analysis of Safety

The Safety Analysis Set will be used for all safety summaries. Summaries will be tabulated by cumulative dose group and for all groups combined.


## 8.6.1. Medical History

The reasons for receiving oliceridine will be summarized by the number and percentage of patients from each initial setting, specialty, and ICD-10 category for each cumulative dose group and for all groups combined using the Safety Analysis Set.

Other medical history collected will be summarized by the number and percentage of patients from each body system and medical condition for each cumulative dose group and for all groups combined using the Safety Analysis Set. All medical hisotry events will be coded using MedDRA version 19.0

Data listing including all medical history regardless of whether or not it was the reason for receiving oliceridine will be produced.

#### 8.6.2. Extent of Exposure and Compliance to Study Treatment

#### 8.6.2.1. Extent of Exposure

Each exposure summary will be summarized for each cumulative dose group and for all groups combined using the Safety Analysis Set.

The method of administration will be summarized by the number and percentage of patients using each method. Patients will have the method of administration categorized as PCA if they received at least 1 PCA dosing. Otherwise the method of administration will be categorized as bolus. Then, regardless of the method of administration, the duration of exposure to study medication will be displayed by summary statistics (mean, standard deviation, median, minimum, and maximum). This duration will be computed as the difference in total hours from the start of the first dose of study medication to the end-time for the last dose of study medication administration.

The total amount of oliceridine administered will be computed regardless of the method of administration within the windows defined in Section 6.2.4. Subsequently, the total amount of oliceridine administered to patients over these periods will be summarized (mean, standard deviation, median, minimum, and maximum) by summary statistics.

Exposure summaries will be repeated by sex, age grouping 1, age grouping 2, race, median baseline NPRS score, BMI, CYP2D6 metabolizer status and initial setting subgroups.

Exposure data including the date, time, method of administration, dose in mg for each administration of oliceridine and the cumulative dose will be listed for each patient.

Boxplots for each cumulative dose and dose duration will be generated by site. A scatterplot will also be generated depicting all patient by duration of treatment and cumulative oliceridine dose.


## 8.6.2.2. Measurements of Treatment Compliance

Treatment consists of parenteral opioid therapy administered by qualified medical personnel. There is no opportunity for self-administration outside of the confines of PCA, and the study drug is not dispensed to an enrolled patient outside of the confines of the investigative site. No summaries of compliance will be performed.

### 8.6.3. Adverse Events

The MedDRA version 19.0 will be used to classify all verbatim AE terms with respect to SOC and PT. Summaries will include only TEAEs and will be summarized for the Safety Analysis Set for each cumulative dose group and for all groups combined.

An overall summary of TEAEs will be performed with the following categories: any TEAE, serious TEAEs, TEAEs with the outcome of fatal, and TEAEs leading to early discontinuation. Severity rating and relationship to study medication categories will also be summarized. The summary will include unique patient counts and percentages based on the number of patients in the cumulative dose group, and the total event count. Overall summary of TEAEs will be repeated by sex, age grouping 1, age grouping 2, race, median baseline NPRS score, BMI, CYP2D6 metabolizer status and initial setting subgroups.

The number and percentage of patients with TEAEs for each cumulative dose group and overall will also be displayed by SOC and PT and will be repeated by BMI and CYP2D6 metabolizer status subgroups. These 3 summary tables will also be repeated for serious TEAEs and TEAEs leading to early discontinuation.

TEAEs will also be summarized by PT only. This summary table will be repeated y BMI and CYP2D6 metabolizer status subgroups.

TEAEs, serious TEAEs and TEAEs resulting in early discontinuation will be summarized by cumulative dose and cumulative time based on the time point intervals defined in section 6.2.4. TEAEs by cumulative dose and cumulative time based on the time point intervals will also be summarized by PTs.

A summary of most common TEAEs will be presented, where PTs occurring in at least 5% of the all treated patients group will be included. Summaries will be sorted by PT in descending frequency in the all treated patients column.

Summaries of TEAEs by maximum severity (mild, moderate, or severe) will be performed by SOC and PT. Patients with missing severities will be counted as severe. Summaries of TEAEs by maximum relationship will be performed by SOC and PT. Patients with missing relationship will be counted as probably related.

The denominator for percentages will be the number of patient within the cumulative dose group for the Safety Analysis Set. The total number of events will be presented


Client: Trevena, Inc. Protocol/CIP #: CP130-3003


along with the patient count and percentage. For summaries by SOC and PT, SOCs will be sorted alphabetically. For summaries only by PT, the sort will be by descending frequency in the all treated patients column. PTs with the same frequency count will be sorted alphabetically.

AE data including start/end time, intensity, any action taken, outcome and whether or not it's serious will be listed for each patient by cumulative dose groups. Lastly, scatterplots will be generated depicting patients' cumulative dose by duration of treatment for patients with at least 1 TEAE, patients with at least 1 related TEAE, patients with at least 1 TEAE leading to early discontinuation and patients with at least 1 SAE.

No statistical inference testing between the treatments will be performed for AEs.

## 8.6.4. Clinical Laboratory Evaluations

All clinical laboratory evaluations will be summarized for the Safety Analysis Set for each cumulative dose group and for all groups combined. Descriptive summaries (mean, SD, median, minimum, and maximum) of absolute values and changes from baseline values will be presented for clinical laboratory values at each time point. Summaries will be performed using the standard units for each analyte. These summaries will be conducted over time using the windows specified in Section 6.2.4.

The number of patients with clinical laboratory values below, within, or above normal ranges for each time point will be tabulated (shift tables) for each clinical laboratory analyte by cumulative dose group.

The proportion of patients who have a clinically significant laboratory result will be summarized by time point for each parameter using frequencies and percentages.

Specific liver-related laboratory results will be summarized by cumulative dose groups and by time point. The specific results summarized will be AST  $\geq$  3 x ULN, ALT  $\geq$  3 x ULN, and AST or ALT  $\geq$  5 x ULN, ALT  $\geq$  5 x ULN, and AST or ALT  $\geq$  5 x ULN; and BILI  $\geq$  2 x ULN.

For clinically significant and shift summaries, the worst overall value reported will displayed. These "worst" results will be calculated as the maximum absolute change from baseline.

In addition, laboratory measurements listing will be presented for each patient.

No statistical inference between the treatments will be performed for laboratory evaluations.


## 8.6.5. Vital Signs

All vital signs will be summarized for the Safety Analysis Set for each cumulative dose group and for all groups combined. Descriptive summaries (mean, SD, median, minimum, and maximum) of actual values and changes from baseline values for systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), respiratory rate (RR), and oxygen saturation will be presented at each time point defined in Section 6.2.4.

Patients meeting the PCSA criterion value or change relative to baseline will be summarized for the Safety Analysis Set for each cumulative dose group and for all groups combined also.

In addition, a listing of each vital signs parameter will be presented for each patient.

## 8.6.6. Physical Examination

Patient listings of whether physical examination was performed or not will be presented for the Safety Analysis Set.

#### 8.6.7.ECG

Continuous descriptive summaries (n, mean, SD, median, minimum, and maximum) of actual values and changes from baseline will be calculated for HR, PR interval, RR interval, QRS interval, QT interval, and QTcF interval for the Safety Analysis Set. These summaries will be provided by time point in accordance with the windoing defined in Section 6.2.4.

The number and percentage of patients with normal and abnormal ECG results will be displayed by each cumulative dose group and for all groups combined.

In addition, a listing of electrocardiogram results will be presented for each patient.

#### **8.6.8.** Subjective Opiate Withdrawal Scale (SOWS)

SOWS total score will be summarized with descriptive statistics (number of patients [N], mean, standard deviation [SD], median, minimum, and maximum) for the Safety Analysis Set. All SOWS results will also be listed by treatment.

#### 8.6.9. Pharmacokinetic Procedures

Plasma concentration values (scheduled and unscheduled) will be summarized for the Safety Analysis Set over time using descriptive summary statistics and the analysis windows described in section 6.2.4. All plasma concentration values will be listed at each time point where an assessment has occurred.


#### 8.7 Analysis of Efficacy Parameters

The Efficacy Analysis Set will be the population for all efficacy variables. Descriptive summary statistics will be tabulated by time interval, by cumulative dose group and for all groups combined. No formal statistical testing will be performed on the efficacy endpoints.

### 8.7.1. Analysis of NPRS

Continuous descriptive summaries (n, mean, SD, median, minimum, and maximum) of actual values and changes from baseline will be calculated for the NPRS values for the Efficacy Analysis Set. All NPRS assessments will be listed for each actual time point where an assessment has occurred.

## 8.7.2. Exploratory Analyses

No exploratory analyses of efficacy data are planned.

#### 9. Computer Software

All analyses will be performed by Chiltern, International, using Version 9.3 or later of SAS® software. All summary tables, figures and data listings will be prepared utilizing SAS® software.

#### 10. REFERENCES

Moline B, R. M. (2012). Validity and Interrater Reliability of the Moline-Roberts Pharmacologic Sedation Scale. *Clinical Nurse Specialist*, 140-148.

<sup>2</sup> Handelsman, L., Cochrane, K., Aronson, M. J. et al. (1987). Two New Rating Scales for Opiate Withdrawal,

American Journal of Alcohol Abuse, 13, 294-308.

<sup>3</sup>McCaffery, M., Beebe, A. (1989) *Pain: Clinical Manual for Nursing Practice* (UK edition). Aylesbury: Mosby.

<sup>4</sup> Pasero, C. (1994). *Acute Pain Service*: Policy and Procedure Manual. Los Angeles, CA: Academy Medical Systems.

## 11. APPENDICES

#### 11.1 APPENDIX 1: VARIABLE DEFINITIONS

Age will be calculated as the informed consent date minus the date of birth divided by 365.25 [Age=(ICF Date-DOB)/365.25].

Body mass index (BMI; kg/m2) is calculated as: weight (kg) / [height (m)]2, rounded to one decimal place.

Client: Trevena, Inc. Protocol/CIP #: CP130-3003


Height and weight are collected in imperial units and will be converted using the following conversion factors:

Height (cm) = height (inches) x 2.54 Weight (kg) = weight (lb) x 0.454

Temperature is collected in degrees Fahrenheit and will be converted to degrees Celcius using the following formula:

Temp (°C) = [temp (°F) – 32] x  $\frac{5}{9}$ 

## **Protocol Number CP130-3003**

A phase 3, multicenter, open-label study to evaluate the safety of oliceridine (TRV130) in patients with acute pain for which parenteral opiod therapy is warranted

Mock Data Displays Final Version 1.0 Date: 20Dec 2016

Prepared for: Trevena, Inc. 1018 West 8<sup>th</sup> Avenue, Suite A King of Prussia, PA 19406

Prepared by: Chiltern International, Inc. 1016 West 9<sup>th</sup> Avenue King of Prussia, PA 19406

This document is confidential information of Trevena. It may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Trevena.

Trevena, Inc.
Protocol CP130-3003
Mock Data Displays

| noon bada biopiajo | |
|---|---|
| Table 14.1.1 Protocol Deviation (Safety Analysis Set) | 6 |
| Table 14.1.2.1 Patient Population (Enrolled Analysis Set) | 8 |
| Table 14.1.2.2 Summary of Safety Analysis Set (Safety Analysis Set) | 9 |
| Table 14.1.2.3 Summary of Reasons for Screen Failure (Enrolled Analysis Set) | 10 |
| Table 14.1.3 Summary of Reasons for Receiving Oliceridine (Safety Analysis Set) | 11 |
| Table 14.1.4 Medical History by Body System and Medical Condition (Safety Analysis Set) | 12 |
| Table 14.1.5 Summary of Patient Disposition (Safety Analysis Set) | 13 |
| Table 14.1.6 Demographic and Baseline Characteristics (Safety Analysis Set) | 14 |
| Table 14.1.7 Summary of Prior Medications by Drug Class and Medication (Safety Analysis Set) | 18 |
| Table 14.1.8 Summary of Concomitant Medications by Drug Class and Medication (Safety Analysis Set) | 19 |
| Table 14.2.1 Summary of Numeric Pain Rating Scale Change From Baseline (Efficacy Analysis Set) | 20 |
| Table 14.3.1.1 Exposure to Study Drug (Safety Analysis Set) | 21 |
| Table 14.3.1.2 Exposure to Study Drug by Sex (Safety Analysis Set) | 22 |
| Table 14.3.1.3 Exposure to Study Drug by Age Group 1 (Safety Analysis Set) | |
| Table 14.3.1.4 Exposure to Study Drug by Age Group 2 (Safety Analysis Set) | 23 |
| Table 14.3.1.5 Exposure to Study Drug by Race (Safety Analysis Set) | 23 |
| Table 14.3.1.6 Exposure to Study Drug by Median Baseline NPRS Score (< Median Baseline NPRS Score , >= Median Baseline NPRS Score) (Safety Analysis Set) | 23 |
| Table 14.3.1.7 Exposure to Study Drug by CYP2D6 Metabolizer Status (Safety Analysis Set) | 23 |
| Table 14.3.1.8 Exposure to Study Drug by BMI Category (Safety Analysis Set) | 23 |
| Table 14.3.1.9 Exposure to Study Drug by Initial Setting (Safety Analysis Set) | 23 |
| Table 14.3.2.1 Summary of Treatment Emergent Adverse Events (TEAE) (Safety Analysis Set) | 24 |
| Table 14.3.2.1.1 Summary of Treatment Emergent Adverse Events (TEAE) by Age Group 1 (Safety Analysis Set) | 26 |
| Table 14.3.2.1.2 Summary of Treatment Emergent Adverse Events (TEAE) by Age Group 2 (Safety Analysis Set) | 26 |
| Table 14.3.2.1.3 Summary of Treatment Emergent Adverse Events (TEAE) by Race (Safety Analysis Set) | 26 |
| Table 14.3.2.1.4 Summary of Treatment Emergent Adverse Events (TEAE) by Median Baseline NPRS Score (< Median Baseline NPRS Score, >= Median Baseline NPRS Score) (Safety Analysis Set) | |
| Table 14.3.2.1.5 Summary of Treatment Emergent Adverse Events (TEAE) by CYP2D6 Metabolizer Status (Safety Analysis Set) | 26 |
| Table 14.3.2.1.6 Summary of Treatment Emergent Adverse Events (TEAE) by BMI Category (Safety Analysis Set) | 26 |
| Table 14.3.2.1.7 Summary of Treatment Emergent Adverse Events (TEAE) by Initial Setting (Safety Analysis Set) | 26 |
| Table 14.3.2.2.1 Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term (Safety Analysis Set) | 27 |

Trevena, Inc.
Protocol CP130-3003
Mock Data Displays

| Table 14.3.2.2.1.1 Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set) |
|---|
| Table 14.3.2.2.1.2 Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by BMI Category (Safety Analysis Set) |
| Table 14.3.2.2.2 Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term (Safety Analysis Set) |
| Table 14.3.2.2.1 Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set) |
| Table 14.3.2.2.2 Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by BMI Category (Safety Analysis Set) |
| Table 14.3.2.2.3 Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term (Safety Analysis Set) |
| Table 14.3.2.2.3.1 Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set) |
| Table 14.3.2.2.3.2 Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term by BMI Category (Safety Analysis Set) |
| Table 14.3.2.3.1 Treatment Emergent Adverse Events (TEAE) in Decreasing Frequency of Preferred Term (Safety Analysis Set) |
| Table 14.3.2.3.1.1 Treatment Emergent Adverse Events (TEAE) in Decreasing Frequency of Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set) |
| Table 14.3.2.3.1.2 Treatment Emergent Adverse Events (TEAE) in Decreasing Frequency of Preferred Term by BMI Category (Safety Analysis Set) |
| Table 14.3.2.4.1 Treatment Emergent Adverse Events (TEAE) by Cumulative Dose and Cumulative Time (Safety Analysis Set) |
| Table 14.3.2.4.2 Serious Treatment Emergent Adverse Events (TEAE) by Preferred Term and Duration of Exposure (Safety Analysis Set) |
| Table 14.3.2.4.3 Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by Preferred Term and Duration of Exposure (Safety Analysis Set) |
| Table 14.3.2.5.1 Treatment Emergent Adverse Events (TEAE) by Cumulative Dose and Cumulative Time by Preferred Term (Safety Analysis Set) |
| Table 14.3.2.6.1 Summary of Most Common Treatment Emergent Adverse Events (>=5% of All Treated Patients) by Decreasing Frequency of Preferred Term (Safety Analysis Set) |
| Table 14.3.2.7.1 Treatment Emergent Adverse (TEAE) by Maximum Severity, System Organ Class and Preferred Term (Safety Analysis Set) |
| Table 14.3.2.8.1 Treatment Emergent Adverse (TEAE) by Maximum Relationship, System Organ Class and Preferred Term (Safety Analysis Set) |
| Table 14.3.3.1 Change from Baseline in Clinical Laboratory Results: Hematology (Safety Analysis Set) |
| Table 14.3.3.2 Summary of Clinical Laboratory Results: Chemistry (Safety Analysis Set) |
| Table 14.3.3.1.1 Clinical Laboratory Hematology Results for Shifts from Baseline (Safety Analysis Set) |
| Table 14.3.3.2.1 Clinical Laboratory Chemistry Results for Shifts from Baseline (Safety Analysis Set) . 41 |

Trevena, Inc. Protocol CP130-3003 Mock Data Displays

| Table 14.3.3.1.2 Clinically Significant Clinical Laboratory Hematology Results (Safety Analysis Set) | 42 |
|---|---|
| Table 14.3.3.2.2 Clinically Significant Clinical Laboratory Chemistry Results (Safety Analysis Set) | 43 |
| Table 14.3.4.1 Select Hepatic Laboratory Findings on Treatment (Safety Analysis Set) | 44 |
| Table 14.3.5.1 Change from Baseline in Vital Signs (Safety Analysis Set) | 45 |
| Table 14.3.5.2 Change from Baseline in Oxygen Saturation (%) (Safety Analysis Set) | 45 |
| Table 14.3.5.1.1 Potentially Clinically Significant Vital Signs | 45 |
| Table 14.3.6.1 Moline-Roberts Pharmacologic Sedation Scale (MRPSS) Total Score at Each Time Pol (Safety Analysis Set) | |
| Table 14.3.7.1 Change from Baseline in Electrocardiogram Results (Safety Analysis Set) | 51 |
| Table 14.3.7.1.1 Selected QTcF Thresholds (Safety Analysis Set) | 53 |
| Table 14.3.7.1.2 Summary of Electrocardiogram (ECG) Findings (Safety Analysis Set) | 54 |
| Table 14.3.8.1 Summary of Subjective Opioid Withdrawal Scale (SOWS) Total Score (Safety Analy Set) | |
| Table 14.3.9.1 Summary of Plasma Concentrations (Safety Analysis Set) | 56 |
| Listing 16.2.1.1 Patient Disposition (Enrolled Analysis Set) | 57 |
| Listing 16.2.1.2 Inclusion/Exclusion Criteria (Enrolled Analysis Set) | 58 |
| Listing 16.2.1.3 Protocol Deviations (Enrolled Analysis Set) | 59 |
| Listing 16.2.2.1 Demographics and Baseline Characteristics (Enrolled Analysis Set) | 60 |
| Listing 16.2.2.2 Prior and Concomitant Medications (Enrolled Analysis Set) | 61 |
| Listing 16.2.2.3 Reason for Receiving Oliceridine (Safety Analysis Set) | 62 |
| Listing 16.2.2.4 Medical History (Enrolled Analysis Set) | 63 |
| Listing 16.2.3.1 Study Drug Administration (Safety Analysis Set) | 64 |
| Listing 16.2.4.1 Numeric Pain Rating Scale (NPRS) Scores (Safety Analysis Set) | 65 |
| Listing 16.2.5.1 Adverse Events (Enrolled Analysis Set) | 66 |
| Listing 16.2.6.1 Vital Signs (Safety Analysis Set) | 67 |
| Listing 16.2.7.1 Laboratory Results: Chemistry (Safety Analysis Set) | 68 |
| Listing 16.2.7.2 Laboratory Results: Hematology (Safety Analysis Set) | 69 |
| Listing 16.2.8 12 Lead Electrocardiogram Results (Safety Analysis Set) | 70 |
| Listing 16.2.9 Subjective Opioid Withdrawal Scale (SOWS) (Safety Analysis Set) | 71 |
| Listing 16.2.10 Physical Examination (Safety Analysis Set) | 72 |
| Listing 16.2.11 Moline-Roberts Pharmacologic Sedation Scale Score (Safety Analysis Set) | 73 |
| Listing 16.2.12.x Patient Profiles for Patients with Durations over 96 Hours (Safety Analysis Set) | 73 |
| Figure 1.1 Duration of Treatment by Site (Safety Analysis Set) | 75 |
| Figure 1.2 Cumulative Dose by Site (Safety Analysis Set) | 76 |
| Figure 2.1 Cumulative Dose by Duration of Treatment (Safety Analysis Set) | 77 |
| Figure 2.1.1 Cumulative Dose by Duration of Treatment for Patients With at Least 1 TEAE (Safety Analysis Set) | 78 |

Trevena, Inc.

Final Version 1.0 20 December 2016

Table 14.1.1
Protocol Deviations
(Safety Analysis Set)

| Protocol Deviation<br>Deviation Criticality | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%)[E] | Oliceridine >4 to 8 mg N=XXX n(%)[E] | Oliceridine >8 to 16 mg N=XXX n(%)[E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>36 mg<br>N=XXX<br>n(%)[E] | All Treated Patients N=XXX n(%)[E] |
|---|---|---|---|---|---|---|
| Number of Patients with<br>a Protocol Deviation | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Procedure Window | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Inclusion/Exclusion<br>Criteria | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Unapproved Medication | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Missed Procedure | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E | ] xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |

Note: E = Number of deviation events.

Percentages are based on the number of patients in each cumulative dose group.


Table 14.1.1(Continued)
 Protocol Deviations
 (Safety Analysis Set)

| Protocol Deviation<br>Deviation Criticality | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>36 mg<br>N=XXX<br>n(%)[E] | All Treated Patients N=XXX n(%)[E] |
|---|---|---|---|---|---|---|
| Informed Consent | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Incorrectly Performed<br>Procedure | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Minor | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |
| Major | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] | xxx (xxx.x)[E] |

Note: E = Number of deviation events.

Percentages are based on the number of patients in each cumulative dose group.


## Table 14.1.2.1 Patient Populations (Enrolled Analysis Set)

| Population | All Enrolled Patients N=XXX n(%) |
|-----------------------|------------------------------------|
| Enrolled Analysis Set | xxx (xxx.x) |
| Safety Analysis Set | xxx (xxx.x) |
| Efficacy Analysis Set | xxx (xxx.x) |

Note: Percentages based on the total number of enrolled patients.


Table 14.1.2.2 Summary of Safety Analysis Set (Safety Analysis Set)

| Population<br>Site Number | Oliceridine <= 4 mg N=XXX n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Safety Analysis Set Site 1 Site 2 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the number of patients in each cumulative dose group.


### Table 14.1.2.3 Summary of Reasons for Screen Failure (Enrolled Analysis Set)

| Parameter | All Enrolled Patients N=XXX n(%) |
|---|---|
| Number of Screen Failure Patients | xxx (xxx.x) |
| Number of Patients with Inclusion Criteria not Met | xxx (xxx.x) |
| Number of Patients not Meeting NPRS of >= 4 | xxx (xxx.x) |
| Number of Patients not Meeting Other Inclusion Criteria | xxx (xxx.x) |
| Number of Patients with Exclusion Criteria Met | xxx (xxx.x) |
| Missing | xxx (xxx.x) |

Note: Percentages based on the total number of enrolled patients.

Patients may fail screening for more than one reason.


Table 14.1.3
Summary of Reasons for Receiving Oliceridine (Safety Analysis Set)

| Initial Setting Specialty ICD-10 Category | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated<br>Patients<br>N=XXX<br>n(%) |
|---|---|---|---|---|---|---|
| Surgical | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <pre><specialty 1=""></specialty></pre> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <icd-10 category=""></icd-10> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <specialty 2=""></specialty> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Medical | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <specialty 1=""></specialty> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <icd-10 category=""></icd-10> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <specialty 2=""></specialty> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ED | | | | | | |
| <specialty 1=""></specialty> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <icd-10 category=""></icd-10> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <specialty 2=""></specialty> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the number of patients in each cumulative dose group.

Patient are only counted in the category if finding is the reason for patient's participation in the study.

Programmers Note: Sort by initial setting (Surg, Med then ED) and by decreasing frequency(all treated patients column) of ICD-10 category.


Table 14.1.4

Medical History by Body System and Medical Condition
(Safety Analysis Set)

| Body System<br>Medical Condition | Oliceridine<br><= 4 mg<br>N=XXX<br>n (%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n (%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n (%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n (%) | Oliceridine<br>>36 mg<br>N=XXX<br>n (%) | All Treated<br>Patients<br>N=XXX<br>n (%) |
|---|---|---|---|---|---|---|
| Number of Patients with at Least 1<br>Medical History | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <body 1="" system=""></body> | | | | | | |
| <condition 1=""></condition> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <condition n=""></condition> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <body 2="" system=""></body> | | | | | | |
| <condition 1=""></condition> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <condition n=""></condition> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | | | | | | |

Note: All medical history events were coded using MedDRA version 19.0.

Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each body system and condition within each cumulative dose group.

Programmer's Note: Order System Organ Class alphabetically and preferred term alphabetically within each SOC. If SOC wraps to a new page, it should be repeated in each page. Sort UNCODED as fist SOC.


### Table 14.1.5 Summary of Patient Disposition (Safety Analysis Set)

| Disposition | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated<br>Patients<br>N=XXX<br>n(%) |
|---|---|---|---|---|---|---|
| Number of Patients That Completed the Study [a] | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Number of Patients That<br>Discontinued Early from Study | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Reason for Early Discontinuation from Study | | | | | | |
| ADVERSE EVENT | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| LACK OF EFFICACY | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| LOST TO FOLLOW-UP | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Study Window of Early Discontinuation [b] | | | | | | |
| <t30 minutes=""></t30> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t2 hours=""></t2> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t96 hours=""></t96> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the number of patients in each cumulative dose group.

- [a] Because the duration of treatment for each patient in this study will be determined by the clinical need for parenteral opioid therapy, a patient will be considered to be a completer if no early termination reason is indicated.
- [b] Study window is defined as the date and time of termination date and time of the first dose of oliceridine. See section 6.2.3 of the SAP for windowed time point intervals.


### Table 14.1.6 Demographic and Baseline Characteristics (Safety Analysis Set)

| Characteristic | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Initial Setting, n(%) | | | | | | |
| Surgical | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Medical | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Emergency Department | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Gender, n(%) | | | | | | |
| Male | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Female | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Age (Years) | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | XXX | XXX | XXX | XXX | XXX |
| Age Group 1 (Years), n(%) | | | | | | |
| < Median | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| >= Median | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the total number of non-missing values in each cumulative dose group.

<sup>[</sup>a] Extensive Metabolizer = Normal functional levels of CYP2D6 in the liver. Poor Metabolizer = Low functional levels of CYP2D6 in the liver.


### Table 14.1.6 (continued) Demographic and Baseline Characteristics (Safety Analysis Set)

| Characteristic | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Age Group 2 (Years), n(%) | | | | | | |
| < 65 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| >= 65 to < 75 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| >= 75 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Race, n(%) | | | | | | |
| <race 1=""></race> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <race n=""></race> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Race Group, n(%) | | | | | | |
| White | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Non-White | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Ethnicity, n(%) | | | | | | |
| <ethnicity 1=""></ethnicity> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <ethnicity n=""></ethnicity> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| CYP2D6 Metabolizer Status [a], n(%) | | | | | | |
| Extensive Metabolizer | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Poor Metabolizer | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the total number of non-missing values in each cumulative dose group.

<sup>[</sup>a] Extensive Metabolizer = Normal functional levels of CYP2D6 in the liver. Poor Metabolizer = Low functional levels of CYP2D6 in the liver.


#### Table 14.1.6 (continued) Demographic and Baseline Characteristics (Safety Analysis Set)

| Characteristic | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Height (cm) | | | | | | |
| N | xxx | XXX | XXX | XXX | XXX | Xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | XXX | XXX | xxx | XXX | Xxx |
| Weight (kg) | | | | | | |
| N | xxx | xxx | XXX | XXX | XXX | Xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | XXX | XXX | XXX | XXX | Xxx |
| BMI (kg/m**2) | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | Xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | XXX | xxx | XXX | XXX | Xxx |
| BMI Group (kg/m**2), n(%) | | | | | | |
| < 25 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| >= 25 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the total number of non-missing values in each cumulative dose group.

<sup>[</sup>a] Extensive Metabolizer = Normal functional levels of CYP2D6 in the liver. Poor Metabolizer = Low functional levels of CYP2D6 in the liver.


#### Table 14.1.6 (continued) Demographic and Baseline Characteristics (Safety Analysis Set)

| Characteristic | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Baseline Pain Intensity | xxx | xxx | xxx | xxx | xxx | Xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | xxx | xxx | xxx | XXX | Xxx |

Note: Percentages are based on the total number of non-missing values in each cumulative dose group.

<sup>[</sup>a] Extensive Metabolizer = Normal functional levels of CYP2D6 in the liver. Poor Metabolizer = Low functional levels of CYP2D6 in the liver.


Table 14.1.7

Summary of Prior Medications by Drug Class and Medication (Safety Analysis Set)

| Drug Class Preferred Name[a] | Oliceridine <= 4 mg N=XXX n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Number of Patients Receiving<br>a Prior Medication | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <class 1=""></class> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred 1=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred n=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <class n=""></class> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred 1=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred n=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each drug class and preferred name within each cumulative dose group.

[a] All medications were coded using WHO DRUG version Mar 1 2016.


Table 14.1.8

Summary of Concomitant Medications by Drug Class and Medication (Safety Analysis Set)

| Drug Class Preferred Name[a] | | iceridine<br><= 4 mg<br>N=XXX<br>n(%) | - | liceridine 4 to 8 mg N=XXX n(%) | | iceridine 8 to 16 mg N=XXX n(%) | | liceridine<br>6 to 36 mg<br>N=XXX<br>n(%) | ( | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | | Treated atients N=XXX n(%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of Patients Receiving a Concomitant Medication | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| <class 1=""></class> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | xxx | (xxx.x) | XXX | (xxx.x) |
| <preferred 1=""></preferred> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| • • • | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| <preferred n=""></preferred> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| <class n=""></class> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| <preferred 1=""></preferred> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| • • • | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |
| <preferred n=""></preferred> | XXX | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) | xxx | (xxx.x) | XXX | (xxx.x) | XXX | (xxx.x) |

Note: Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each drug class and preferred name within each cumulative dose group.

[a] All medications were coded using WHO DRUG version Mar 1 2016.


Table 14.2.1

Summary of Numeric Pain Rating Scale Change From Baseline (Efficacy Analysis Set)

| Windowed<br>Time Point [a] | Baseline/<br>Observed/<br>Change from<br>Baseline | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|---|
| Baseline [b] | | | | | | | |
| N | Observed | xxx | XXX | xxx | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | xxx | XXX | xxx | XXX | XXX | XXX |
| <t30 minutes=""></t30> | | | | | | | |
| N | Baseline[c] | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Missing | | xxx | XXX | xxx | XXX | XXX | XXX |
| N | Observed | xxx | xxx | xxx | xxx | xxx | xxx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | XXX | XXX | XXX | XXX | XXX | XXX |
| N | Change | XXX | XXX | XXX | XXX | XXX | xxx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | XXX | XXX | XXX | XXX | XXX | XXX |

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

<sup>[</sup>c] Only patients with both a baseline value and a windowed time point value are summarized at a given windowed time point.


### Table 14.3.1.1 Exposure to Study Drug (Safety Analysis Set)

| | Oliceridine<br><=4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>> 36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Method of Administration, n(%) | | | | | | |
| Bolus | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| PCA | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Exposure to Oliceridine [a] (Hours) | | | | | | |
| N | Xxx | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| Number of Patients Exposed by Study Window [b], n(%) | | | | | | |
| <t30 minutes=""></t30> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ••• | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t96 hours=""></t96> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Cumulative Oliceridine Dose (mg) | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX |

Note: Percentages are based on the number of patients in each cumulative dose group.

<sup>[</sup>a] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.

<sup>[</sup>b] See section 6.2.3 of the SAP for windowed time point intervals.


### Table 14.3.1.2 Exposure to Study Drug by Sex (Safety Analysis Set)

| | Oliceridine<br><=4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>> 36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Sex: Male | xxx | xxx | xxx | xxx | xxx | xxx |
| Method of Administration, n(%) | | | | | | |
| Bolus | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| PCA | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Exposure to Oliceridine [a] (Hours) | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| Number of Patients Exposed by Study Window [b], n(%) | | ( | ( | ( | ( | |
| <t30 minutes=""></t30> | , | , | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x |
| · · · | xxx (xxx.x) | , | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x |
| <t96 hours=""></t96> | XXX (XXX.X) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x |
| Cumulative Oliceridine Dose (mg) | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Sex: Female | xxx | XXX | XXX | XXX | xxx | xxx |

Note: Percentages are based on the number of patients in each cumulative dose group.

<sup>[</sup>a] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.

<sup>[</sup>b] See section 6.2.3 of the SAP for windowed time point intervals.


#### Use the same template as for Table 14.3.1.2 for the following tables:

Table 14.3.1.3

Exposure to Study Drug by Age Group 1 (Safety Analysis Set)

Table 14.3.1.4

Exposure to Study Drug by Age Group 2 (Safety Analysis Set)

Table 14.3.1.5

Exposure to Study Drug by Race (Safety Analysis Set)

Table 14.3.1.6

Exposure to Study Drug by Median Baseline NPRS Score (< Median Baseline NPRS Score , >= Median Baseline NPRS Score) (Safety Analysis Set)

Table 14.3.1.7

Exposure to Study Drug by CYP2D6 Metabolizer Status (Safety Analysis Set)

Table 14.3.1.8

Exposure to Study Drug by BMI Category (Safety Analysis Set)

Table 14.3.1.9

Exposure to Study Drug by Initial Setting (Safety Analysis Set)

Trevena, Inc.

Protocol CP130-3003


Page x of y

Table 14.3.2.1
Summary of Treatment Emergent Adverse Events (TEAE)
(Safety Analysis Set)

| | Oliceridine<br><=4 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>> 36 mg<br>N=XXX<br>n(%)[E] | All Treated Patients N=XXX n(%)[E] |
|---|---|---|---|---|---|---|
| Patients with at Least 1 TEAE | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] |
| Patient with at Least 1 Serious<br>TEAE | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |
| Number of Patients Who Had a TEAE with a Fatal Outcome | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |
| Patients with at Least 1 TEAE<br>Leading to Early Study Medication<br>Discontinuation [a] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] |
| Due to Study Medication-Related TEAE [b] | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) [xxx] | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Due to Serious TEAE | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] |
| Patients with TEAEs by Maximum<br>Severity | | | | | | |
| Mild | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] |
| Moderate | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| Severe[c] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group.

All adverse events were coded using MedDRA version 19.0. TEAEs are defined in section 6.3.3 of the SAP.

- [a] AE recorded as having an action taken of drug discontinued.
- [b] Includes events recorded as possibly related, probably related, or missing.
- [c] Missing severities are assumed to be severe.
- [d] Missing relationships are assumed to be probably related.


#### Table 14.3.2.1(continued) Summary of Treatment Emergent Adverse Events (TEAE) (Safety Analysis Set)

| | Oliceridine<br><=4 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%)[E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%)[E] | Oliceridine > 36 mg N=XXX n(%)[E] | All Treated Patients N=XXX n(%)[E] |
|---|---|---|---|---|---|---|
| Patients with TEAEs by Maximum | | | | | | |
| Not Related | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| Unlikely Related | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| Possibly Related | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| Probably Related | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| Possibly or Probably Related | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group.

All adverse events were coded using MedDRA version 19.0. TEAEs are defined in section 6.3.3 of the SAP.

- [a] AE recorded as having an action taken of drug discontinued.
- [b] Includes events recorded as possibly related, probably related, or missing.
- [c] Missing severities are assumed to be severe.
- [d] Missing relationships are assumed to be probably related.


#### Use the same template as for Table 14.3.2.1 for the following tables:

Table 14.3.2.1.1

Summary of Treatment Emergent Adverse Events (TEAE) by Age Group 1 (Safety Analysis Set)

Table 14.3.2.1.2

Summary of Treatment Emergent Adverse Events (TEAE) by Age Group 2 (Safety Analysis Set)

Table 14.3.2.1.3

Summary of Treatment Emergent Adverse Events (TEAE) by Race (Safety Analysis Set)

Table 14.3.2.1.4

Summary of Treatment Emergent Adverse Events (TEAE) by Median Baseline NPRS Score (< Median Baseline NPRS Score , >= Median Baseline NPRS Score)

(Safety Analysis Set)

Table 14.3.2.1.5

Summary of Treatment Emergent Adverse Events (TEAE) by CYP2D6 Metabolizer Status (Safety Analysis Set)

Table 14.3.2.1.6

Summary of Treatment Emergent Adverse Events (TEAE) by BMI Category (Safety Analysis Set)

Table 14.3.2.1.7

Summary of Treatment Emergent Adverse Events (TEAE) by Initial Setting (Safety Analysis Set)


| System Organ Class<br>Preferred Term | Oliceridine <= 4 mg N=XXX n(%) [E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) [E] | Oliceridine >36 mg N=XXX n(%) [E] | All Treated Patients N=XXX n(%) [E] |
|---|---|---|---|---|---|---|
| Patients with at Least 1 TEAE | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] |
| <soc 1=""></soc> | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <preferred 1="" term=""></preferred> | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| ••• | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <preferred n="" term=""></preferred> | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <soc n=""></soc> | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <preferred 1="" term=""></preferred> | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| ••• | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <preferred n="" term=""></preferred> | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |

Note: E = Number of events.

All adverse event terms were coded using MedDRA dictionary version 19.0.

Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each system organ class and each preferred term.

TEAEs are defined in section 6.3.3 of the SAP.

Source: Listing x.x.x Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm


#### Use the same template as for Table 14.3.2.2.1 for the following tables:

Table 14.3.2.2.1.1

Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set)

Table 14.3.2.2.1.2

Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by BMI Category (Safety Analysis Set)

Table 14.3.2.2.2

Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term (Safety Analysis Set)

Table 14.3.2.2.2.1

Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set)

Table 14.3.2.2.2.2

Serious Treatment Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term by BMI Category (Safety Analysis Set)

Table 14.3.2.2.3

Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term (Safety Analysis Set)

Table 14.3.2.2.3.1

Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term by

CYP2D6 Metabolizer Status

(Safety Analysis Set)

Table 14.3.2.2.3.2

Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by System Organ Class and Preferred Term by
BMI Category
(Safety Analysis Set)


| Preferred Term | Oliceridine <= 4 mg N=XXX n(%) [E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) [E] | All Treated Patients N=XXX n(%) [E] |
|---|---|---|---|---|---|---|
| Patients with at Least 1 TEAE | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |
| <preferred 1="" term=""></preferred> | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] |
| <preferred 2="" term=""></preferred> | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| ••• | | | | | | |
| <preferred n="" term=""></preferred> | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |

Note: E = Number of events.

All adverse event terms were coded using MedDRA dictionary version 19.0.

Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each preferred term.

TEAEs are defined in section 6.3.3 of the SAP.

Preferred terms are sorted in descending patient level incidence in the All Treated Patients column.

Programmer's Note: Order preferred terms based on the All Treated Patients column. If preferred terms have the same patient count, order by descending event count and then alphabetically.


#### Use the same template as for Table 14.3.2.3.2 for the following tables:

Table 14.3.2.3.1.1

Treatment Emergent Adverse Events (TEAE) in Decreasing Frequency of Preferred Term by CYP2D6 Metabolizer Status (Safety Analysis Set)

Table 14.3.2.3.1.2

Treatment Emergent Adverse Events (TEAE) in Decreasing Frequency of Preferred Term by BMI Category (Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm


#### Table 14.3.2.4.1 Treatment Emergent Adverse Events (TEAE) by Cumulative Dose and Cumulative Time (Safety Analysis Set)

| Cumulative<br>Duration of<br>Exposure[a] | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) [E] | All Treated Patients N=XXX n(%) [E] |
|---|---|---|---|---|---|---|
| Patients with at<br>Least 1 TEAE | xxx (xxx.x)[xxx] | xxx (xxx.x)[xxx] | xxx (xxx.x)[xxx] | xxx (xxx.x)[xxx] | xxx (xxx.x)[xxx] | xxx (xxx.x) [xxx] |
| <t30 minutes=""> <t2 hours=""></t2></t30> | xxx (xxx.x)[xxx] | xxx (xxx.x)[xxx] | xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx]<br>xxx (xxx.x) [xxx] |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group and cumulative duration of exposure windowed time point. The denominators for each cell can be referenced in table 14.3.1.1.

See section 6.2.3 of the SAP for windowed time point intervals.

TEAEs are defined in section 6.3.3 of the SAP.

[a] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.


#### Use the same template as for Table 14.3.2.4.1 for the following tables:

Table 14.3.2.4.2

Serious Treatment Emergent Adverse Events (TEAE) by Preferred Term and Duration of Exposure (Safety Analysis Set)

Table 14.3.2.4.3

Treatment Emergent Adverse Events (TEAE) Resulting in Early Discontinuation by Preferred Term and Duration of Exposure (Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm

Trevena, Inc.

Protocol CP130-3003


Page x of y

Table 14.3.2.5.1

Treatment Emergent Adverse Events (TEAE) by Cumulative Dose and Cumulative Time by Preferred Term (Safety Analysis Set)

| Preferred Term [a] Cumulative Duration of Exposure[b] | Oliceridine | Oliceridine | Oliceridine | Oliceridine | Oliceridine | All Treated |
|---|---|---|---|---|---|---|
| | <= 4 mg | >4 to 8 mg | >8 to 16 mg | >16 to 36 mg | >36 mg | Patients |
| | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX |
| | n(%) [E] | n(%) [E] | n(%) [E] | n(%) [E] | n(%) [E] | n(%) [E] |
| <preferred 1="" term=""> <t30 minutes=""> <t2 hours=""></t2></t30></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred 2="" term=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <preferred n="" term=""></preferred> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group and cumulative duration of exposure windowed time point. The denominators for each cell can be referenced in table 14.3.1.1.

Patients are counted once within each preferred term.

See section 6.2.3 of the SAP for windowed time point intervals.

TEAEs are defined in section 6.3.3 of the SAP.

[a] All adverse event terms were coded using MedDRA dictionary version 19.0.

[b] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.


# Table 14.3.2.6.1 Summary of Most Common Treatment Emergent Adverse Events (>=5% of All Treated Patients) by Decreasing Frequency of Preferred Term (Safety Analysis Set)

| Preferred Term[a] | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) [E] | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) [E] | All Treated Patients N=XXX n(%) [E] |
|---|---|---|---|---|---|---|
| Patients with at Least 1 TEAE | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] |
| <preferred 1="" term=""></preferred> | xxx (xxx.x)<br>[xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] | xxx (xxx.x) [xxx] |
| <preferred n="" term=""></preferred> | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] | xxx (xxx.x)<br>[xxx] |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each preferred term.

TEAEs are defined in section 6.3.3 of the SAP.

Preferred terms are sorted in descending patient level incidence in the All Treated Patients column.

[a] All adverse event terms were coded using MedDRA dictionary version 19.0.

Programmer's Note: Order preferred terms based on the All Treated Patients column. If preferred terms have the same patient count, order by descending event count and then alphabetically.


Table 14.3.2.7.1

Treatment Emergent Adverse (TEAE) by Maximum Severity, System Organ Class and Preferred Term (Safety Analysis Set)

| System Organ Class<br>Preferred Term[a]<br>Severity | | liceridine<br><= 4 mg<br>N=XXX<br>n(%) [E] | > | liceridine<br>4 to 8 mg<br>N=XXX<br>n(%) [E] | > | liceridine<br>8 to 16 mg<br>N=XXX<br>n(%) [E] | - | liceridine<br>16 to 36 mg<br>N=XXX<br>n(%) [E] | 0 | Dliceridine<br>>36 mg<br>N=XXX<br>n(%) [E] | A | ll Treated<br>Patients<br>N=XXX<br>n(%) [E] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patients with at<br>Least 1 TEAE | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] |
| Mild | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Moderate | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Severe | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] |
| <soc 1=""></soc> | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] |
| Mild | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Moderate | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Severe | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| <preferred 1="" term=""></preferred> | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Mild | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Moderate | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| Severe | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] |
| ••• | | | | | | | | | | | | |

Note: E = Number of events.

Percentages are based on the number of patients in each cumulative dose group.

Patients are counted once within each system organ class and preferred term.

TEAEs are defined in section 6.3.3 of the SAP.

If a patient had more than one occurrence of the same event, the highest severity is summarized. Missing severities are assumed to be severe.

[a] All adverse event terms were coded using MedDRA dictionary version 19.0.

Programmer's Note: Order system organ class alphabetically and preferred term alphabetically withing each system organ class. Repeat SOC on each page if it wraps on to multiple pages.


### Table 14.3.2.8.1 Treatment Emergent Adverse (TEAE) by Maximum Relationship, System Organ Class and Preferred Term (Safety Analysis Set)

| System Organ Class<br>Preferred Term[a]<br>Relationship | | | | | | | | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) [E] | | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) [E] | | ll Treated Patients N=XXX n(%) [E] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patients with at<br>Least 1 TEAE | xxx | (xxx.x) [xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | xxx | (xxx.x)[xxx |
| Not Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Unlikely Related | | (xxx.x)[xxx] | | | | | | | | | | · - |
| Possibly Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Probably Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Possibly or Probably Related [b] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| <pre><soc 1=""></soc></pre> | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Not Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx |
| Unlikely Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Possibly Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Probably Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Possibly or Probably<br>Related [b] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| <preferred 1="" term=""></preferred> | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | xxx | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x) [xxx] | XXX | (xxx.x)[xxx |
| Not Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Unlikely Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Possibly Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Probably Related | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |
| Possibly or<br>Probably<br>Related [b] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx] | XXX | (xxx.x)[xxx |

Note: E = Number of events.


Percentages are based on the number of patients in each cumulative dose group. Patients are counted once within each system organ class and preferred term. TEAEs are defined in section 6.3.3 of the SAP.

- [a] All adverse event terms were coded using MedDRA dictionary version 19.0.
- [b] Missing relationships are assumed to be probably related.

Programmer's Note: Order system organ class alphabetically and preferred term alphabetically withing each system organ class. Repeat SOC on each page if it wraps on to multiple pages.

Source: Listing x.x.x
Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm


### Table 14.3.3.1 Change from Baseline in Clinical Laboratory Results: Hematology (Safety Analysis Set)

| Parameter (unit)<br>Windowed Time Point[a] | Baseline/<br>Observed/<br>Change from<br>Baseline | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|---|
| <parameter (unit)="" x=""></parameter> | | | | | | | |
| Baseline[b] | | | | | | | |
| n | Observed | XXX | XXX | xxx | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX |
| <t30 minutes=""></t30> | | | | | | | |
| n | Baseline[c] | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| n | Observed | xxx | xxx | xxx | xxx | xxx | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| n | Change | xxx | xxx | xxx | xxx | xxx | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |

Note: Percentages are based on the number of patients in each cumulative dose group.

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

Trevena, Inc.

Protocol CP130-3003

Page x of y

| Parameter (unit) | Baseline/ | Oliceridine | Oliceridine | Oliceridine | Oliceridine | Oliceridine | All Treated |
|---|---|---|---|---|---|---|---|
| | Observed/ | <= 4 mg | >4 to 8 mg | >8 to 16 mg | >16 to 36 mg | >36 mg | Patients |
| | Change from | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX |
| Windowed Time Point[a] | Baseline | 14 212121 | 14 212121 | 14 212121 | 14 212121 | 14 212121 | 14 212121 |

<sup>[</sup>c] Only patients with both a baseline value and a windowed time point value are summarized at a given windowed time point.

Programmer's Note: Repeat Parameter (unit) in each page if it wraps on to multiple pages.

Use the same template as for Table 14.3.3.1 for the following tables:

Table 14.3.3.2

Summary of Clinical Laboratory Results: Chemistry (Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm


Table 14.3.3.1.1
Clinical Laboratory Hematology Results for Shifts from Baseline (Safety Analysis Set)

| | | | | | Post Baseline | | |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | | | Low | Normal | High - | Total | Missing |
| Windowed Time Point[a] | Cumulative dose group | Baseline<br>[b] | n (%) | n (%) | n (%) | n (%) | _ |
| <parameter (unit)="" 1=""></parameter> | Oliceridine <= 4 mg (N=XXX) | | | | | | |
| Worst Post Baseline | | Low | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | High | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Total | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Missing | xxx | XXX | xxx | XXX | XXX |
| <t30 minutes=""></t30> | | Low | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | High | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Total | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Missing | XXX | XXX | XXX | XXX | XXX |
| <time n="" point=""></time> | | Low | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx |
| .110 101110 11 | | Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | High | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Total | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | XXX |
| | | Missing | XXX | XXX | XXX | XXX | XXX |

Note: Low = below normal reference range; Normal = within normal reference range; High = above normal reference range.

Percentages are based on the number of patients with a non-missing baseline and post-baseline windowed time point value within each windowed time point, parameter and cumulative dose group.

Worst post-baseline is calculated as the most extreme absolute change from baseline value.

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.


Use the same template as for Table 14.3.4.1.3 for the following tables:

Table 14.3.3.2.1
Clinical Laboratory Chemistry Results for Shifts from Baseline (Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx

Data Extraction: yyyymmdd Output Date: yyyymmddthh:mm

## Table 14.3.3.1.2 Clinically Significant Clinical Laboratory Hematology Results (Safety Analysis Set)

| Parameter (unit) Windowed Time Point [a] Interpretation | Oliceridine <= 4 mg N=XXX n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Patients with at Least 1 Clinically<br>Significant Hematology Result | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <parameter (unit)="" 1=""></parameter> | | | | | | |
| Baseline[b] | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, NCS | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, CSig | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Worst Post-Baseline Value | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, NCS | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, CSig | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t30 minutes=""></t30> | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, NCS | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, CSig | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: NCS = Not clinically significant; CSig = Clinically significant.

Clinical significance is based on the investigator interpretation as recorded.

Percentages are based on the number of patients with a non-missing baseline and post-baseline windowed time point value within each windowed time point, parameter and cumulative dose group.

Worst post-baseline is calculated as the most extreme absolute change from baseline value.

Trevena, Inc.

Protocol CP130-3003

Page x of y

[a] See section 6.2.3 of the SAP for windowed time point intervals.

[b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

Programmer's Note: Continue with all parameters and all windowed time points even if all counts are 0.

Use the same template as for Table 14.3.3.1.2 for the following tables:

Table 14.3.3.2.2
Clinically Significant Clinical Laboratory Chemistry Results
(Safety Analysis Set)

Source: Listing x.x.x Program Name: s<nnn>xxxx


# Table 14.3.4.1 Select Hepatic Laboratory Findings on Treatment (Safety Analysis Set)

| Windowed Time Point [a] Test Result | Oliceridine <= 4 mg N=XXX n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Patients with at Least 1 Hepatic<br>Laboratory Finding | | | | | | |
| AST >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ALT >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| AST or ALT >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| AST >=5 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ALT >=5 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| AST or ALT >=5 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| BILI >=2 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t30 minutes=""></t30> | | | | | | |
| AST >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| ALT >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| AST or ALT >=3 X ULN | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: ALT = Alanine Aminotransferase; AST = Asparate Aminotransferase; BILI = Total Bilirubin; ULN = Upper Limit of Normal.

Percentages are based on the number of patients with a non-missing windowed time point value within each windowed time point and cumulative dose group.

[a] See section 6.2.3 of the SAP for windowed time point intervals.

Programmer's Note: Continue with all windowed time points and criteria rows, even if all counts are 0..

Source: Listing x.x.x Program Name: s<nnn>xxxx

. . .


## Table 14.3.5.1 Change from Baseline in Vital Signs (Safety Analysis Set)

| Parameter (unit)<br>Windowed Time Point[a] | Baseline/<br>Observed/<br>Change from<br>Baseline | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|---|
| <parameter (unit)="" x=""></parameter> | | | | | | | |
| Baseline[b] | | | | | | | |
| n | Observed | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| <t30 minutes=""></t30> | | | | | | | |
| n | Baseline[c] | XXX | XXX | xxx | XXX | XXX | xxx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| n | Observed | xxx | xxx | xxx | xxx | xxx | xxx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |
| n | Change | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |

[a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

<sup>[</sup>c] Only patients with both a baseline value and a windowed time point value are summarized at a given windowed time point. *Programmer's Note: Repeat Parameter (unit) in each page if it wraps on to multiple pages.* 


# Table 14.3.5.2 Change from Baseline in Oxygen Saturation (%) (Safety Analysis Set)

| Windowed Time Point[a] | Baseline/<br>Observed/<br>Change from Baseline | <= 4 mg | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|---|
| Baseline[b] | | | | | | | |
| n | Observed | xxx | xxx | xxx | xxx | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| <t30 minutes=""></t30> | | | | | | | |
| n | Baseline[c] | XXX | XXX | xxx | xxx | xxx | xxx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| n | Observed | XXX | XXX | xxx | xxx | xxx | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| n | Change | XXX | XXX | xxx | xxx | XXX | XXX |
| Mean (SD) | <u> </u> | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Min, Max | | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |

[a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

<sup>[</sup>c] Only patients with both a baseline value and a windowed time point value are summarized at a given windowed time point.


Table 14.3.5.1.1
Potentially Clinically Significant Vital Signs (Safety Analysis Set)

| PCSA Criterion | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Systolic Blood Pressure <= 80 mmHg | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Systolic Blood Pressure >= 180 mmHg | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Systolic Blood Pressure change from baseline > 25% increase | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Systolic Blood Pressure change from baseline > 25% decrease | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Diastolic Blood Pressure <= 40 mmHg | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Diastolic Blood Pressure >= 110 mmHg | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |

Note: Percentages are based on the number of patients in each cumulative dose group.

Trevena, Inc.
Protocol CP130-3003

Page x of y

# Table 14.3.5.1.1(continued) Potentially Clinically Significant Vital Signs (Safety Analysis Set)

| PCSA Criterion | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| Diastolic Blood Pressure change from baseline > 25% increase | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Diastolic Blood Pressure<br>change from baseline<br>> 25% decrease | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Pulse Rate <= 40 bpm | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Pulse Rate >= 120 bpm | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Pulse Rate change from baseline > 15 bpm increase | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |
| Pulse Rate change from baseline > 15 bpm Decrease | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |

Note: Percentages are based on the number of patients in each cumulative dose group.


# Table 14.3.5.1.1(continued) Potentially Clinically Significant Vital Signs (Safety Analysis Set)

| PCSA Criterion | Oliceridine | Oliceridine | Oliceridine | Oliceridine | Oliceridine | All Treated |
|---|---|---|---|---|---|---|
| | <= 4 mg | >4 to 8 mg | >8 to 16 mg | >16 to 36 mg | >36 mg | Patients |
| | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX | N=XXX |
| Oxygen Saturation < 90% | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) | xxx (xxx.x%) |

Note: Percentages are based on the number of patients in each cumulative dose group.


Table 14.3.6.1

Moline-Roberts Pharmacologic Sedation Scale (MRPSS) Total Score at Each Time Point (Safety Analysis Set)

| Windowed Time Point [a]<br>Sedation | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated<br>Patients<br>N=XXX<br>n(%) |
|---|---|---|---|---|---|---|
| <baseline [b]=""></baseline> | | | | | | |
| 1. None to Minimal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 2. Anxiolysis | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 3. Moderate Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 4. Moderate Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 5. Deep Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 6. General Anesthesia | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t30 minutes=""></t30> | | | | | | |
| 1. None to Minimal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 2. Anxiolysis | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 3. Moderate Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 4. Moderate Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x |
| 5. Deep Sedation | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| 6. General Anesthesia | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x |

. . .

Note: Percentages are based on the number of patients in each cumulative dose group.

Somnolence/sedation was measured with the Moline-Roberts Pharmacologic Sedation Scale (MRPSS).

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.

<sup>[</sup>b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.


# Table 14.3.7.1 Change from Baseline in Electrocardiogram Results (Safety Analysis Set)

| Parameter (unit)<br>Windowed Time Point [a] | Baseline/<br>Observed/<br>Change from<br>Baseline | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|---|
| <pre><parameter (unit)="" x=""> Baseline [b]</parameter></pre> | | | | | | | |
| n | Observed | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | XXX | XXX | XXX | XXX | XXX | XXX |
| <t30 minutes=""></t30> | | | | | | | |
| n | Baseline [c] | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | XXX | XXX | xxx | xxx | xxx | XXX |
| n | Observed | XXX | XXX | xxx | xxx | xxx | XXX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | | XXX | XXX | xxx | xxx | xxx | XXX |
| n | Change | XXX | XXX | xxx | xxx | xxx | xxx |
| Mean (SD) | - | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Missing | | XXX | XXX | XXX | XXX | XXX | XXX |

Note: Percentages are based on the number of patients in each cumulative dose group.

Trevena, Inc.

Protocol CP130-3003


Page x of y

- [a] See section 6.2.3 of the SAP for windowed time point intervals.
- [b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.
- [c] Only patients with both a baseline value and a windowed time point value are summarized at a given windowed time point.

Programmer's Note: Repeat Parameter (unit) in each page if it wraps on to multiple pages.

Source: Listing x.x.x
Program Name: s<nnn>xxxx


## Table 14.3.7.1.1 Selected QTcF Thresholds (Safety Analysis Set)

| Windowed Time Point [a] | Oliceridine <= 4 mg N=XXX n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Overall | xxx | xxx | xxx | xxx | xxx | xxx |
| Change from Baseline of > 30 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Change from Baseline of > 60 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Increase to > 500 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t30 minutes=""></t30> | xxx | xxx | XXX | xxx | XXX | xxx |
| Change from Baseline of > 30 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Change from Baseline of > 60 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Increase to > 500 msec | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| • • • | | | | | | |

Note: Percentages are based on the number of patients in each cumulative dose group.

Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.

[a] See section 6.2.3 of the SAP for windowed time point intervals.

Programmer's Note: Display all ECG windowed time points after overall.


Table 14.3.7.1.2

Summary of Electrocardiogram (ECG) Findings (Safety Analysis Set)

| Windowed Time Point [a]<br>Finding | Oliceridine<br><= 4 mg<br>N=XXX<br>n(%) | Oliceridine<br>>4 to 8 mg<br>N=XXX<br>n(%) | Oliceridine<br>>8 to 16 mg<br>N=XXX<br>n(%) | Oliceridine<br>>16 to 36 mg<br>N=XXX<br>n(%) | Oliceridine<br>>36 mg<br>N=XXX<br>n(%) | All Treated Patients N=XXX n(%) |
|---|---|---|---|---|---|---|
| Patients with at Least 1 Clinically<br>Significant ECG Result | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Baseline [b] | | | | | | |
| Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, NCS | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, CSig | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| <t30 minutes=""></t30> | | | | | | |
| Normal | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, NCS | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Abnormal, CSig | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Missing | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |

Note: NCS = Not clinically significant; CSig = Clinically significant.

Clinical significance is based on the investigator interpretation as recorded.

Percentages are based on the number of patients in each cumulative dose group.

- [a] See section 6.2.3 of the SAP for windowed time point intervals.
- [b] Baseline is the last non-missing value prior to the patient receiving the first dose of oliceridine.


Table 14.3.8.1
Summary of Subjective Opioid Withdrawal Scale (SOWS) Total Score (Safety Analysis Set)

| | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| N | XXX | xxx | xxx | xxx | xxx | xxx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Missing | XXX | XXX | XXX | XXX | XXX | XXX |

Note: Total score is derived by summing the individual symptom intensities. If no more than half of the symptoms are missing, imputation with the mean score of the non-missing questions is used to calculate total score. If more than half of the symptoms are missing the total score is also set to missing.


# Table 14.3.9.1 Summary of Plasma Concentrations (Safety Analysis Set)

| Windowed Time Point[a] | Oliceridine<br><= 4 mg<br>N=XXX | Oliceridine<br>>4 to 8 mg<br>N=XXX | Oliceridine<br>>8 to 16 mg<br>N=XXX | Oliceridine<br>>16 to 36 mg<br>N=XXX | Oliceridine<br>>36 mg<br>N=XXX | All Treated<br>Patients<br>N=XXX |
|---|---|---|---|---|---|---|
| T30 Minutes | | | | | | |
| N | xxx | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | XXX | XXX | XXX | xxx | xxx | XXX |
| T1.5 Hours | | | | | | |
| N | xxx | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Missing | xxx | xxx | xxx | xxx | xxx | XXX |

Note: Unscheduled PK samples will be displayed in the listing.

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.

Sex/Age/

Group

Cumulative Dose

Trevena, Inc.
Protocol CP130-3003

Patient ID


Listing 16.2.1.1
Patient Disposition
(Enrolled Analysis Set)

Exposure [b])

Date/Time of End
of Treatment
(Cumulative Date of Study Primary Reason for
Duration of Completion/ Termination

Discontinuation[a]

(Other)

[a] Date/time of study completion/discontinuation is the date collected at the end of study instead of the of the date/time last dose received.

Date/Time of

Oliceridine

First Dose of

<sup>[</sup>b] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.


Listing 16.2.1.2
Inclusion/Exclusion Criteria
(Enrolled Analysis Set)

Sex/Age/

Patient ID Cumulative Dose Group Met all Eligibility Criteria? Criteria not Met

Note: Patients may fail screening for more than one reason.


Listing 16.2.1.3
Protocol Deviations
(Enrolled Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Patient ID/Sex/Age Deviation Type Deviation Text Detail Deviation Criticality IRB Reportable?/Report Date

Note: IRB = Institutional Review Board.

Source: Listing x.x.x
Program Name: s<nnn>xxxx


#### Listing 16.2.2.1 Demographics and Baseline Characteristics (Enrolled Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

| | | | Baseline | | | |
|---|---|---|---|---|---|---|
| | | Informed | Height (cm)/ | | | CYP2D6 |
| Patient | Race/ | Consent | Weight (kg)/ | ASA Physical Status | ESI | Phenotype |
| ID/Sex/Age | Specify Ethnicity | Date | BMI (kg/m^2) | Classificiation [a] | Classification | (EM vs PM) |

Note: BMI = Body mass index; ASA = American Society of Anesthesiologists; ESI = Emergency Severity Index; EM = Extensive metabolizer; PM = Poor metabolizer.

- [a] ASA Physical Status is defined as follows: I Normal healthy patient; II Patient with mild systemic disease; III Patient with severe systemic disease; IV Patient with severe systemic disease that is a constant threat to life; V Moribund patient who is not expected to survive without the operation; VI Declared brain-dead patient whose organs are being removed for donor purposes.
- [b] Extensive Metabolizer patients include those with a predictive phenotype of Ultra Metabolizer or Extensive Metabolizer; Poor Metabolizer patients include those with a predictive phenotype of Intermediate Metabolizer or Poor Metabolizer.


Listing 16.2.2.2
Prior and Concomitant Medications
(Enrolled Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

| | Base Preferred Name/ | | Stop | | Dose | | | | Given |
|---|---|---|---|---|---|---|---|---|---|
| Patient | ATC Class/ | Start | Date/Time | | and | Route | | | for AE?/ |
| ID/Sex/Age | Medication | Date/Time | or Ongoing | P/C | Unit | (Other) | Frequency | Indication | AE # |

Note: AE = Adverse Event; ATC = Anatomic Theraputic Chemical; P = Prior Medication; C = Concomitant Medication;

Programmer's Note: Sort by Start date/time. For missing date/times sort alphabetically


Listing 16.2.2.3
Reason for Receiving Oliceridine
(Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Patient ID/Sex/Age Initial Setting Condition ICD-10 Code/ICD Description Specialty

Source: Listing x.x.x
Program Name: s<nnn>xxxx


Listing 16.2.2.4 Medical History (Enrolled Analysis Set)

| | Sex/Age/ | | | | | |
|---|---|---|---|---|---|---|
| | Cumulative | Medical | System Organ | | | Stop Date or |
| Patient ID | Dose Group | History | Class | Preferred Term | Start Date | Ongoing |


Listing 16.2.3.1
Study Drug Administration
(Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Start Windowed Time
Patient ID/Sex/Age Method of Administration Date/Time Point [a] Dose Received Cumulative Dose

Note: Asterisk (\*) denotes the last dose received.
[a] See section 6.2.3 of the SAP for windowed time point intervals.


Listing 16.2.4.1
Numeric Pain Rating Scale (NPRS) Scores
(Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Patient ID/Sex/Age Assessment Date/Time Windowed Time Point[a] Numeric Pain Rating Scale (NPRS) Score

Note: Asterisk (\*) denotes the value used in descriptive summary statistics. [a] See section 6.2.3 of the SAP for windowed time point intervals.

Source: Listing x.x.x Program Name: s<nnn>xxxx


Listing 16.2.5.1 Adverse Events (Enrolled Analysis Set)

Patient ID/Sex/Age/Cumulative Dose Group: 1001/Male/30/ Oliceridine <= 4 mg

Start

System Organ Class/ Date/Time/

Concomitant Preferred Term [a]/ End Date/Time Intenity/ medication

Action Serious?/ Additional Verbatim Term Reason for Serious Information AE # (or Ongoing) Relationship given?/CM # Taken Outcome

Note: All adverse events were coded using MedDRA version 19.0. TEAEs are defined in section 6.3.3 of the SAP.

Source: Listing x.x.x Program Name: s<nnn>xxxx


Listing 16.2.6.1 Vital Signs (Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

| Collecti<br>Patient ID/Sex/Age Date/Tir | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Respiratory<br>Rate<br>(breaths/min) | Temperature | Pulse<br>Oximetry<br>(SpO2 %) |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

Note: Asterisk (\*) denotes the value used in descriptive summary statistics.

Source: Listing x.x.x
Program Name: s<nnn>xxxx

<sup>[</sup>a] See section 6.2.3 of the SAP for windowed time point intervals.


Listing 16.2.7.1
Laboratory Results: Chemistry
(Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Lab Collection Windowed Time Lab Test
Patient ID/Sex/Age Date/Time Point [a] (Unit) Lab Value Overall Interpretation

Note: N = Normal; NCS = Not Clinically Significant; Csig = Clinically Significant; Asterisk (\*) denotes the value used in descriptive summary statistics.

The investigator will exercise his or her medical and scientific judgement in deciding whether an abnormal laboratory finding is clinically significant.

[a] See section 6.2.3 of the SAP for windowed time point intervals.

Source: Listing x.x.x
Program Name: s<nnn>xxxx


Use the same template as for Listing 16.2.7.1 for the following listings:

Listing 16.2.7.2
Laboratory Results: Hematology
(Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx


# Listing 16.2.8 12 Lead Electrocardiogram Results (Safety Analysis Set)

Patient ID/Sex/Age/Cumulative Dose Group: 1001/Male/30/ Oliceridine <= 4 mg

| | Windowed | | | RR | QRS | QT | QTcF | | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment<br>Date/Time | Time<br>Point[a] | Heart Rate (beats/min) | PR Interval (msec) | Interval (msec) | Interval (msec) | Interval (msec) | Interval (msec) | Interpreta<br>tion | Abnormal,<br>Sepcify |

Note: Csig = Clinically Significant; NCS = Not Clinically Significant.

Asterisk (\*) denotes the value used in descriptive summary statistics.

Source: Listing x.x.x
Program Name: s<nnn>xxxx


Listing 16.2.9
Subjective Opioid Withdrawal Scale (SOWS)
(Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Assessment

Patient ID/Sex/Age Date/Time

Symptom

Intensity Rating [a]

[a] 0 = Not at all; 1 = A little; 2 = Moderately; 3 = Quite a bit; 4 = Extremely.

Source: Listing x.x.x Program Name: s<nnn>xxxx


Listing 16.2.10 Physical Examination (Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Patient ID/Sex/Age

Assessment Date/Time

Changes From Previous Visit?

Source: Listing x.x.x
Program Name: s<nnn>xxxx


Listing 16.2.11
Moline-Roberts Pharmacologic Sedation Scale Score (Safety Analysis Set)

Cumulative Dose Group: Oliceridine <= 4 mg

Patient ID/Sex/Age Assessment Date/Time Windowed Time Point [a] Total Score

Note: Asterisk (\*) denotes the value used in descriptive summary statistics.

[a] See section 6.2.3 of the SAP for windowed time point intervals.

Source: Listing x.x.x
Program Name: s<nnn>xxxx


#### Listing 16.2.12.x Patient Profiles for Patients with Durations Over 96 Hours (Safety Analysis Set)

Patient ID/Sex/Age/Cumulative Dose Group: xxxxx

Cumulative Duration of Oliceridine Dose Exposure [a] Administration (mg) (Hours) Completed the Study?[b] Reason for Early Termination

xx xx xx xx

| Base Preferred Name/ | | | | Dose | | | | |
|---|---|---|---|---|---|---|---|---|
| ATC Class/ | Start | Stop Date/Time | | and | Route | | | Given for |
| Medication | Date/Time | or Ongoing | P/C | Unit | (Other) | Frequency | Indication | AE?/ AE # |

System Organ Class/
Preferred Term [a]/
Verbatim Term

Start Date/Time/
End Date/Time Intensity/ Action Serious?/
Relationship Taken Outcome Reason for Seriousness

Note: AE = Adverse Event; ATC = Anatomic Theraputic Chemical; P = Prior Medication; C = Concomitant Medication; All adverse events were coded using MedDRA version 19.0.

<sup>[</sup>a] Duration is defined as the difference in total hours from the first dose to the last dose of of study medication.

<sup>[</sup>b] Because the duration of treatment for each patient in this study will be determined by the clinical need for parenteral opioid therapy, a patient will be considered to be a completer if no early termination reason is indicated.

Trevena, Inc.

Protocol CP130-3003

Page x of y

Figure 1.1
Duration of Treatment by Site
(Safety Analysis Set)



[a] Duration is defined as the difference in total hours from the start of the first dose of study medication to end-time for the last dose of study drug administration.

Programmer's Note: Limit to 10 sites per page.

Trevena, Inc.

Protocol CP130-3003


Page x of y

Figure 1.2 Cumulative Dose by Site (Safety Analysis Set)



Programmer's Note: Limit to 10 sites per page.


Figure 2.1
Cumulative Dose by Duration of Treatment
(Safety Analysis Set)



Note: Each dot in the graph represents a patient.

[a] Duration is defined as the difference in total hours from the start of the first dose of study medication to end-time for the last dose of study drug administration.


#### Use the same template as for Figure 2.1 for the following Figures:

Figure 2.1.1

Cumulative Dose by Duration of Treatment for Patients With at Least 1 TEAE (Safety Analysis Set)

Figure 2.1.2

Cumulative Dose by Duration of Treatment for Patients With at Least 1 Related TEAE (Safety Analysis Set)

Figure 2.1.3

Cumulative Dose by Duration of Treatment for Patients With at Least 1 TEAE Leading to Early Discontinuation (Safety Analysis Set)

Figure 2.1.4

Cumulative Dose by Duration of Treatment for Patients With at Least 1 SAE (Safety Analysis Set)

Source: Listing x.x.x
Program Name: s<nnn>xxxx